## Janssen Research & Development

## Statistical Analysis Plan

Prospective, multi-center, single-arm, open-label long-term study assessing the safety, tolerability, and effectiveness of macitentan in Fontan-palliated adult and adolescent subjects

AC-055H302/RUBATO-OL; Phase 3

ACT-064992 / JNJ-67896062 (macitentan)

**Status:** Approved

Date: 17 December 2021

Prepared by: Actelion Pharmaceuticals Ltd., a Janssen Pharmaceutical Company of Johnson &

Johnson

Document No.: EDMS-RIM-265704, 1.0

Compliance: The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

# **TABLE OF CONTENTS**

| TABL | LE OF CONTENTS | 2 |
|---|---|---|
| LIST | OF TABLES | 3 |
| LIST | OF FIGURES | 3 |
| VERS | SION HISTORY | 4 |
| | INTRODUCTION | |
| 1.1. | Objectives and Endpoints | |
| 1.2. | Study Designs | 6 |
| 2. | STATISTICAL HYPOTHESES | 8 |
| 3. | SAMPLE SIZE DETERMINATION | 8 |
| 4. | POPULATIONS (ANALYSIS SETS) FOR ANALYSIS | 8 |
| 5. | STATISTICAL ANALYSES | 10 |
| 5.1. | General Considerations | |
| 5.1.1. | | |
| 5.1.2. | ,,,,,,,,,, | |
| 5.1.2. | | |
| 5.1.2. | | |
| 5.1.2. | | |
| 5.1.2. | | |
| 5.1.2. | | |
| 5.1.2. | | |
| 5.2. | Participant Dispositions | |
| 5.2.1. | , | |
| 5.2.2. | , | |
| 5.2.3. | | |
| 5.3. | Extent of Exposure and Compliance | |
| 5.4. | Safety Analysis | |
| 5.4.1. | | |
| 5.4.2. | | |
| 5.4.3. | | |
| 5.4.4. | | |
| 5.4.4. | | |
| 5.4.4. | | |
| 5.4.5. | 5 1 7 | |
| 5.5. | Efficacy Analysis | |
| 5.5.1. | | |
| 5.5.2.<br>5.5.3. | | |
| 5.5.s.<br>5.6. | · | |
| 5.6.1.<br>5.6.1. | Other Analyses Definition of Subgroups and subgroup analyses | 30 |
| | SUPPORTING DOCUMENTATION | |
| 6.1. | Appendix 1: List of Abbreviations | |
| 6.2. | Appendix 2: Changes to Protocol-Planned Analyses | |
| 6.3. | Appendix 3: Demographic and Baseline Characteristics | |
| 6.3.1. | | |
| 6.3.2. | | |
| 6.4. | Appendix 4: Protocol Deviations and Quality Tolerance Limits (QTL) | 42 |

| 6.5. Ar | opendix 5: Prior and Concomitant Medications | 49 |
|---|---|---|
| | Prior Medications | |
| | Concomitant Medications | |
| | Concomitant Medications at Start of Study Treatment in Analysis Set | |
| 6.6. Ap | ppendix 6: Intervention Compliance | 51 |
| 6.7. A | ppendix 7: Adverse Events of Special Interest and COVID-19 related AEs | 52 |
| 7. REF | ERENCES | 53 |
| LIST OF | TABLES | |
| Table 1: | SAP Version History Summary | 4 |
| Table 2: | Study Documents. | 5 |
| Table 3: | Analysis Set Definitions | |
| Table 4: | Usage of Analysis Sets | |
| Table 5: | Time Windows for the OL Period and Day 30 FU | |
| Table 6: | Thresholds for Marked Laboratory Abnormalities | |
| Table 7: | Table of Subgroups for Analyses | |
| Table 8: | Demographic Variables | |
| Table 9: | Baseline Disease Characteristics | |
| Table 10: | PD Classification Based on AC-055H302 (RUBATO OL) | |
| Table 11: | Quality Tolerance Limits as per Integrated Analytical Risk-Based Monitoring Plan | 48 |
| LIST OF | FIGURES | |
| Figure 1: | RUBATO OL Study Design | 6 |
| Figure 2: | RUBATO OL Study Design (with S-FU in the AC-055H301 RUBATO DB Study) | 7 |

# **VERSION HISTORY**

**Table 1:** SAP Version History Summary

| SAP Version | Approval Date | Change | Rationale |
|-------------|------------------|----------------|-----------------|
| 1 | 17 December 2021 | Not Applicable | Initial release |

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) describes in detail the methods, conduct and content of the data analysis of AC-055H302/RUBATO open-label extension study (hereafter referred to as the RUBATO OL study) for the purpose of the abbreviated Clinical Study Report (CSR). As planned in the protocol, some of the analyses are based on data pooled with data from the corresponding core study, AC-055H301/RUBATO (hereafter referred to as the RUBATO DB study).

Following the evaluation of the study results from the RUBATO DB study, a sponsor decision was taken to terminate the RUBATO OL study early. For this reason, an abbreviated CSR is planned. All safety data and selected non-safety data obtained will be summarized in the abbreviated CSR.

All analyses are exploratory in nature and therefore no multiplicity issues are foreseen.

This SAP refers to the documents listed in Table 2.

#### **Table 2:** Study Documents

| Document | Date, Version |
|---|---|
| Study Protocol AC-055H302 (RUBATO OL) | Final Version 4 (D-20.426) |
| Study Protocol AC-055H301 (RUBATO) | Final Version 10 (D-20.425) |
| AC-055H301 SAP for clinical study report (CSR) | Final Version 5 (EDMS-RIM-264216, 3.0) |
| AC-055H301 SDTM annotated eCRF specifications | Version 1.0, 8 September 2021, or latest implemented version |
| AC-055H302 SDTM annotated eCRF specifications | Version 11.0 (draft 19 October 2021), or latest implemented version |
| Study Protocol AC-055H302 (RUBATO OL) COVID-19<br>Appendix | Approved version, 17 June 2020 (D-20.159) |
| Study Protocol AC-055H301 (RUBATO) COVID-19 Appendix | Approved version, 17 June 2020 (D-20.158) |

Source data for the AC-055H301/RUBATO DB will be Analysis Data Model (ADaM) data sets derived for the AC-055H301/RUBATO CSR SAP. Except where otherwise specified, all definitions and conventions used in the CSR SAP of this study will be applied, as applicable.

Source data for the RUBATO OL study are provided as Statistical Analysis Software (SAS®) data sets according to Clinical Data Interchange Standards Consortium Study Data Tabulation Model (SDTM). Source data are provided according to the Database Release Plan document.

The pooling of RUBATO DB and RUBATO OL means that the data from the same subjects randomized in RUBATO DB will be concatenated with their data from the OL study. The concatenation of data from the same subject is referred to as 'pooling' in this document.

### 1.1. Objectives and Endpoints

The primary objective of the study is to assess the long-term safety and tolerability of macitentan in Fontan-palliated adult and adolescent subjects. This SAP describes how safety and selected

efficacy will be analyzed and summarized in order to support the abbreviated RUBATO OL CSR. This includes the concatenation of data from studies RUBATO DB and RUBATO OL.

## 1.2. Study Designs

RUBATO DB is a prospective, multi-center, double-blind, randomized, placebo controlled, parallel-group Phase 3 study assessing the efficacy and safety of macitentan in Fontan-palliated adult and adolescent subjects.

At least 134 subjects were to be randomized in a 1:1 ratio to receive 52 weeks of treatment with either macitentan or placebo. Randomization was stratified by geographical region (America, Europe, Asia, Oceania). The study was to be conducted in approximately 31 investigational sites in 11 countries.

The study is completed, database was locked on 02-Sep-2021.

RUBATO OL is a prospective, multi-center, single-arm, open-label, long-term, Phase 3 study assessing the safety, tolerability, and effectiveness of macitentan in Fontan-palliated adult and adolescent subjects. The overall study design of RUBATO OL is depicted in Figure 1.

Figure 1: RUBATO OL Study Design



DB = Double-blind (study); EOS = End-of-Study; EOT = End-of-Treatment; OL = Open-label (extension); V = visit = Telephone call (for visit).

In instances where administration of RUBATO OL study treatment does not immediately follow End-of-Treatment (EOT) in the RUBATO DB study, the subject will enter the DB S-FU period per protocol until administration of the first dose of the OL study treatment occurs (Figure 2).

OL enrollment AC-055H301 RUBATO AC-055H302 RUBATO OL Macitentan 10 mg Macitentan 10 mg Every 26 Placebo weeks until study FOT weeks 26 Safety Safety Treatment (blinded) Treatment (Open-label) Follow-up Follow-up 30 days 30 days **DB Randomization** DB EOT **DB EOS EOS** Visits: V1 V2 V3 EOT

Figure 2: RUBATO OL Study Design (with S-FU in the AC-055H301 RUBATO DB Study)

DB = Double-blind (study); EOS = End-of-Study; EOT = End-of-Treatment; OL = Open-label (extension); S-FU = Safety Follow-up; V = visit; = Telephone call (for visit).

No S-FU will be performed for subjects entering a post-trial access program at individual subject's EOT for the RUBATO OL study.

Visit and assessment schedules of the RUBATO DB and the RUBATO OL studies can be found in the corresponding protocols.

As it was recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of the clinical studies, the sponsor issued Study Protocol COVID-19 Appendices to provide options for study related subject management in the event of disruption to the conduct of the study. Discontinuations of study interventions and withdrawal from the study were to be documented with the prefix "COVID-19-related" in the electronic case report form (eCRF). Also, protocol deviations (PDs) linked to COVID-19, were to be prefixed with the text "COVID-19 related" in the clinical database.

The RUBATO DB results showed no clinically meaningful difference favoring macitentan 10 mg that would provide treatment benefit to Fontan-palliated patients, and therefore, the sponsor has decided that the RUBATO OL study will be terminated early.

### 2. STATISTICAL HYPOTHESES

No formal hypothesis testing is performed. All efficacy analyses are purely descriptive.

### 3. SAMPLE SIZE DETERMINATION

Not applicable. RUBATO OL is an extension study of the RUBATO DB study, hence the sample size of the pools will be up to the number of randomized subjects in the RUBATO DB study, with no sample size statistical considerations.

# 4. POPULATIONS (ANALYSIS SETS) FOR ANALYSIS

Table 3 below describes analysis sets, periods and treatment arms used.

**Table 3:** Analysis Set Definitions

| Analysis Set | Period definition | Treatment Arms |
|---|---|---|
| RUBATO Open-label | The RUBATO Open-label Extension Set (OLES) includes | DB-Placebo |
| Extension Set (OLES) | all subjects treated with macitentan in RUBATO OL study. | DB-Macitentan 10 |
| | Only data from the OL period (as defined in Section 5.1.2.6) | mg |
| | are considered with the exception of baseline data | OL Macitentan 10 |
| | (including demographic data, medical and disease history | mg (All OLES |
| | data, prior medication) which may origin from the DB | subjects) |
| | period. Treatment arms "DB-Macitentan 10 mg" and "DB- | |
| | Placebo" follow the treatment arm from RUBATO DB | |
| | safety set (SS), i.e., are based on actual treatment received | |
| | in study RUBATO DB. | |
| RUBATO pool (FAS and | Pool of all RUBATO DB and RUBATO OL data. Data | Placebo/Macitentan |
| SS) | from the same subjects randomized in DB are concatenated | 10 mg (Plc/Maci) |
| | with their data from the OL extension study. Baseline is | |
| | defined relative to first intake of study medication in the | |
| | RUBATO DB study, as defined in the RUBATO DB study | |
| | SAP. Treatment arms for FAS follow the treatment arm | |
| | assignment from RUBATO DB FAS analyses, i.e., | |
| | treatment as randomized. | 3.6 10 |
| | Treatment arms for SS follow the treatment arm assignment | Macitentan 10 mg |
| | from RUBATO DB SS analyses, i.e., are based on actual | /Macitentan 10 mg |
| | treatment received in study RUBATO DB. | (Maci/Maci) |
| RUBATO Total | Only subjects receiving at least one dose of macitentan | Macitentan 10 mg |
| Macitentan Analysis Set | (either in RUBATO DB or RUBATO OL) are included. | Pool |
| (TMAS) (SS) | Only subjects from the macitentan arm in the RUBATO DB | |
| | SS analyses are considered to have received macitentan in | |
| | the RUBATO DB, their data are concatenated with their | |
| | data from the OL extension. For subjects from the DB study | |
| | SS placebo arm, only data with assessment dates during the | |
| | OL period (as defined in in Section 5.1.2.6) are considered, with the exception of baseline data (including demographic | |
| | data, medical and disease history data, prior medication) | |
| | which may origin from the DB period. Baseline is defined | |
| | relative to first intake of macitentan study treatment (either | |
| | in RUBATO DB or RUBATO OL). | |

FAS – Full analysis set, SS – Safety Set.

# Table 4 describes usage of analysis sets.

**Table 4:** Usage of Analysis Sets

| | Analysis Set | | |
|---|---|---|---|
| Endpoint | RUBATO<br>OLES | RUBATO pool | RUBATO<br>TMAS (SS) |
| Efficacy | | | |
| CPET (peak VO <sub>2</sub> , VO <sub>2</sub> at VAT) | Yes | Yes (FAS) | |
| PA-Ac (Mean count per minute) | Yes | Yes (FAS) | |
| Fontan-palliated clinical worsening | | Yes (FAS) | |
| Fontan-palliated morbidity | | Yes (FAS) | |
| Safety | | | |
| AEs (incl SAEs, AESI, AE by intensity, by relationship, AE leading to study treatment discontinuation, fatal AEs) | Yes | Yes (SS) for<br>Maci/Maci Arm<br>only | Yes |
| Death | | Yes (SS) | |
| Vital signs (BP, pulse) including peripheral oxygen saturation (SpO <sub>2</sub> ) and body weight, over time | Yes | Yes (SS) | |
| Systolic blood pressure outlier analyses | Yes | Yes (SS) for<br>Maci/Maci Arm<br>only | Yes |
| Laboratory results, over time | Yes | Yes (SS) | |
| Marked laboratory abnormalities/laboratory outlier analyses | Yes | Yes (SS) for<br>Maci/Maci Arm<br>only | Yes |
| Echocardiography numerical results, over time | Yes | Yes (SS) | |
| Echocardiography valvular defects | Yes | Yes (SS) | Yes |
| Exposure/Compliance | Yes | Yes (SS) | Yes |
| Demographics | Yes | | Yes |
| Baseline Disease Characteristics | Yes | | Yes |
| Disposition | Yes | | Yes |
| Protocol Deviations | Yes | | |
| Concomitant Medications | Yes | | Yes |

#### 5. STATISTICAL ANALYSES

#### 5.1. General Considerations

SAS (Statistical Analysis System®) version 9.4 is used for all the statistical analyses, except if otherwise specified.

Data will be listed and summarized by appropriate descriptive statistics (tables or figures).

General rules for data presentations as described below are followed unless otherwise specified:

- All listings will be sorted by treatment arm, site ID, subject ID and when appropriate by visit / date of assessment. All data collected will be displayed, including unscheduled visits (if any).
- In summary tables, treatment arms will be presented in columns from left to right following the order shown in Table 3.
- If on a table or figure a visit/timepoint is empty (i.e., zero subjects across all treatment arms), this visit/timepoint is not displayed.

#### 5.1.1. Visit Windows

As subjects do not always adhere to the protocol visit schedule, the following rules are applied to assign actual visits to analysis visits.

Visit-based analyses are planned to be conducted based on the RUBATO OLES and on the RUBATO pool. Analysis visits for the RUBATO DB period within the RUBATO pool follow the RUBATO DB SAP, visits labelled "Baseline" or "Week xx" in the RUBATO DB CSR SAP are re-labelled to "DB Baseline" or "DB Week xx". For the RUBATO OL period, analyses visits are assigned according to Table 5.

Safety assessments are generally reported based on the nominal visit, i.e., according to the visit reported in the database, however for subjects who discontinued OL study treatment prematurely with available premature EOT visit, the EOT assessments may be re-assigned to a scheduled visit according to the windows specified in Table 5 in case the premature EOT visit assessment is treatment emergent (i.e., within 30 days after study treatment discontinuation).

All efficacy assessments (including unscheduled ones) are assigned to analysis visits as follows: If a subject has two or more assessments in one visit window, the assessment closest to the target day will be used as the analysis visit for that visit window. The other additional assessment(s) will not be used in by-visit summaries or analyses, but they can be used for determination of other endpoints (e.g., time to event endpoints). If two assessments are equidistant from the target day within a visit window, the later visit is used. If more than one value falls on the same timepoint then the one with the worst assessment (i.e., lowest peak VO<sub>2</sub>, VO<sub>2</sub> at VAT, PA-Ac mean count per minute) is used. All assignments will be made in chronological order. Once an assessment is assigned to a visit window, it will no longer be used for a later time point.

Assessments which fall outside of any planned window will not be included in by-visit summary tables and graphs but will be included in outlier tables and into individual subject listings.

| Parameter | Analysis Visit<br>(label on output) | Time Interval (OL Day)* | Target Time<br>Point<br>(OL Day) |
|---|---|---|---|
| PA-Ac | OL Baseline | 1 to 30 | 2-10 |
| Efficacy parameters. | OL Week 26 | 92 to 273 | 183 |
| Safety parameters (for EOT | OL Week 52 | 274 to 455 | 365 |
| visit remapping only) | OL Week 78 | 456 to 637 | 547 |
| | OL Week 104 | 638 to 819 | 729 |
| | OL Week 130 | 820 to 1001 | 911 |
| | OL Week 156 | 1002 to 1183 | 1093 |
| Laboratory (aminotransferases | Day 30 FU | ≥ Analysis<br>Set FOT + 28 | Analysis Set EOT + |

Table 5: Time Windows for the OL Period and Day 30 FU

## 5.1.2. Definition of Baseline, Periods and Dates/Days

#### 5.1.2.1. Baseline

The **DB** baseline is used as derived in the core DB study (i.e., not re-derived). Except where otherwise specified in the RUBATO DB CSR SAP, DB baseline is defined as the last non-missing assessment obtained before or on the day of the start of study treatment.

The **macitentan baseline** is defined as the last value assessed prior or on the macitentan treatment start date (either in the core RUBATO DB study or in the RUBATO OL extension) defined in Section 5.1.2.2.

**Baseline in OLES** is generally defined as the last non-missing assessment obtained prior or on the RUBATO OL treatment start date defined in Section 5.1.2.2. For PA-Ac, OLES baseline is based on assessments recorded after RUBATO OL treatment start date, details are given in Section 5.5.2.

Baseline in RUBATO pool and RUBATO DB set corresponds to DB baseline.

Baseline in TMAS set corresponds to macitentan baseline.

### 5.1.2.2. Treatment Start Date (Day 1) and Day Numbering in Analysis Sets

The **DB treatment start date (DB Day 1)** is used as derived in the RUBATO DB study (i.e., not re-derived).

The **OL** treatment start date (**OL Day 1**) is the date of first dose of macitentan treatment in the RUBATO OL study. This is the "Treatment start date" (defined as the date the first dose of study treatment intake) from the first interval, in chronological order, recorded in the "Study Drug Log" eCRF module of RUBATO OL.

The macitentan treatment start date (macitentan Day 1), is defined to be the date of first dose of macitentan either in the core RUBATO DB study or in the extension RUBATO OL. For subjects

<sup>\*</sup> Relative to OL Day 1 (defined in Section 5.1.2.2)

from the macitentan group according to the SS in RUBATO DB, it is the DB treatment start date (as defined above), for subjects from the placebo group according to the SS in RUBATO DB it is the OL treatment start (as defined above).

**OLES Day 1** corresponds to OL treatment start date (OL Day 1).

**RUBATO pool Day 1 and RUBATO DB Day 1** set correspond to DB treatment start date (DB Day 1).

**TMAS Day 1** corresponds to macitentan treatment start date (macitentan Day 1).

All safety and efficacy assessments/events (with the exception of Fontan-palliated clinical worsening and Fontan-palliated morbidity) at all visits will be assigned a day relative to analysis set Day 1.

Day or relative day for a visit/ assessments/event is defined as:

- Visit/assessment/event date − Date of analysis set Day 1 + 1, if visit/assessment/event date is ≥ date of analysis set Day 1
- Visit date/assessment/event Date of analysis set Day 1, if visit/assessment/event date < date of analysis set Day 1

There is no 'Day 0'.

Day of Fontan-palliated clinical worsening and Fontan-palliated morbidity in the RUBATO pool is calculated relative to the randomization date:

• Date of Fontan-palliated clinical worsening / morbidity – Randomization Date + 1

### 5.1.2.3. End of Treatment (EOT) Date

**DB EOT** corresponds to study treatment end date as defined in the RUBATO DB CSR SAP.

**OL EOT** is only defined for subjects treated with OL treatment and corresponds to "Treatment end date" from the last interval, in chronological order, recorded in the "Study Drug Log" eCRF form.

**Macitentan EOT** is defined to be the date of last dose of macitentan either in the RUBATO DB study or in the extension RUBATO OL. For subjects from the macitentan group according to the SS RUBATO DB who did not enter the RUBATO OL study, this is the DB EOT (as defined in above), otherwise it is the OL EOT as defined above.

**EOT in OLES** corresponds to OL EOT.

**EOT in RUBATO pool** corresponds to OL EOT for subjects treated with OL treatment, and to DB EOT for subjects not treated with OL treatment.

**EOT in TMAS** corresponds to macitentan EOT.

## 5.1.2.4. End of Study (EOS) Date

**DB EOS** corresponds to EOS date as defined in the RUBATO DB CSR SAP.

**OL EOS** is only defined for subjects treated with OL treatment and corresponds to the date entered on the 'Visit Summary-EOS' eCRF Form. For subjects who died, EOS corresponds to the date of death. If a subject is lost to follow-up, EOS corresponds to the date of last successful contact from the 'Study Discontinuation' eCRF form.

**EOS** in **OLES** corresponds to OL EOS.

**EOS** in RUBATO pool and in TMAS corresponds to OL EOS for subjects treated with OL treatment, and to DB EOS for subjects not treated with OL treatment.

#### 5.1.2.5. **DB Period**

All visits, assessments and events dated prior to the OL treatment start date (as defined in Section 5.1.2.2) are considered to belong to the DB period. For subjects not in the OLES (i.e., those not dosed with OL treatment), all data collected in RUBATO DB database is included and assigned to DB period.

#### 5.1.2.6. **OL Period**

It is the period between OL treatment start date (as defined in Section 5.1.2.2) and OL EOS (as defined in Section 5.1.2.4), limits included.

### 5.2. Participant Dispositions

As per protocol amendment 3 (protocol version 4), RUBATO OL was planned to continue for each subject until the last subject has globally completed 104 weeks (2 years) of treatment. Subjects who enrolled the into RUBATO OL (i.e., were treated with OL treatment) and who did not consent to protocol version 4, but completed 104 weeks of OL treatment and the corresponding S-FU period under protocol version 3, are considered treatment and study completers in the OL period.

The following definitions are relevant to provide the disposition information.

### 5.2.1. Study Treatment Discontinuation

The number and percentage of subjects who discontinued study treatment (incl discontinuation reasons) in the analysis set are presented for the RUBATO OLES and the RUBATO TMAS.

In both studies, study treatment discontinuations are collected in the "Study Drug Log" eCRF form and identified as those with a treatment end date and associated reason ('What was the reason for treatment end?') answered 'Premature Discontinuation'. Reasons for study treatment discontinuation are collected in the "Premature Discontinuation of Study Treatment' eCRF form. The following reasons for permanent treatment discontinuation are displayed (including if documented to be "COVID-19 related" as per prefix in database):

#### Death

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

- Lost to follow-up
- Pre-specified study treatment discontinuation criteria
- Adverse Event (this combines reports of subject and physician decision)
- Lack of Efficacy (this combines reports of subject and physician decision)
- Other
  - Other medical reasons (this combines reports of subject and physician decision)
  - Other non-medical reasons (this combines reports of subject and physician decision)
  - No reason provided (Subject decision)
  - Sponsor decision Study termination
  - Sponsor decision Other

For analyses based on the RUBATO TMAS an additional Study Treatment Discontinuation reason is defined as

• Completed treatment in RUBATO DB study but not enrolled into RUBATO OL study

For the RUBATO OLES, only RUBATO OL eCRF forms are considered whereas for the RUBATO TMAS, information is concatenated from both study eCRFs. For subjects who prematurely discontinued study treatment in the DB study and who entered the OL study after completing the week 52 PTOP visit in the DB study, the study treatment discontinuation reason in DB is not considered for treatment disposition in RUBATO TMAS.

An individual listing of subjects who discontinued study treatment prematurely and related reason(s) will be provided for the RUBATO OLES and the RUBATO TMAS.

### 5.2.2. Study Discontinuation

The number and percentage of subjects who prematurely discontinued study (including discontinuation reasons) in the analysis set is presented for the RUBATO OLES and the RUBATO TMAS.

In both studies, study treatment discontinuations are collected in the "Study Discontinuation" eCRF page.

Subjects who withdrew from the study are those with any withdrawal reason entered in the "Study Discontinuation" eCRF module. The following reasons for study discontinuation are displayed (including if documented to be "COVID-19 related" as per prefix in database):

- Death
- Lost to follow-up
- Adverse Event (this combines reports of subject and physician decision)

- Lack of Efficacy (this combines reports of subject and physician decision)
- Other
  - Other medical reasons (this combines reports of subject and physician decision)
  - Other non-medical reasons (this combines reports of subject and physician decision)
  - No reason provided (Subject decision)
  - Sponsor decision Study termination
  - Sponsor decision Other

For analyses based on the RUBATO TMAS an additional Study Discontinuation reason is defined as:

• Completed DB study but not enrolled into RUBATO OL study

For the RUBATO OLES, only RUBATO OL eCRF forms are considered whereas for the RUBATO TMAS, information is concatenated from both study eCRF and OL disposition overwrites DB disposition.

An individual listing of subjects who discontinued study prematurely and related reason(s) will be provided for the RUBATO OLES and the RUBATO TMAS.

## 5.2.3. Other Disposition Information

For the RUBATO OLES, the study and treatment disposition as defined in the RUBATO DB SAP will be presented to inform on the number of subjects seamlessly entering the RUBATO OL study versus subjects enrolling into OL after entering the DB study PTOP.

In addition, the distribution (number and percentage of subjects) by geographical region, country, and site ID will be presented for the RUBATO OLES and the RUBATO TMAS.

The number of subjects in the different analysis sets will be tabulated and a listing of subject membership in the different analysis sets is provided.

### 5.3. Extent of Exposure and Compliance

Exposure and compliance variables are derived and summarized for the RUBATO OLES, RUBATO pool (SS), and the RUBATO TMAS.

The exposure within an analysis set is evaluated first in terms of study treatment duration, including study treatment interruptions. The study treatment exposure (in days) in analysis set is calculated as:

treatment end date in analysis set -treatment start date in analysis set +1

In addition, the study treatment exposure is evaluated in terms of actual days exposed to study treatment, excluding any temporary interruptions. A subject is considered to have had a study

treatment interruption if the reason for treatment end is either 'Temporarily interrupted due to an AE' or 'Temporarily interrupted not due to an AE' ("Study Drug Log" eCRF form), corresponding treatment end dates, and treatment restart dates are taken from the "Study Drug Log" eCRF form. For the RUBATO pool and the RUBATO TMAS, also gaps between DB EOT (defined in Section 5.1.2.3) and OL treatment start date (defined in Section 5.1.2.2) are considered as interruption. Treatment interruptions and gaps between DB EOT and OL treatment start of more than 30 days are flagged.

The study treatment exposure, excluding any temporary interruptions, is calculated as:

Study treatment exposure in analysis set — total duration of interruptions in analysis set.

Where the total duration of interruptions is the sum of all treatment interruptions. The duration of each treatment interruption is calculated as:

Treatment restart date (or OL start date) – treatment end date (or DB treatment end date) – 1.

Compliance is assessed as a percentage based on exposure as defined above from the study drug log, calculated for each pool as follows:

Study treatment exposure in analysis set excluding interruptions  $\times$  100 Study treatment exposure in analysis set

*Note:* Compliance below 100% must not be indicative of a deviation from the protocol since there are protocol mandated reasons for interruptions and a protocol allowed gap in transition from DB to OL study.

Corresponding categorical variables (not mutually exclusive) are derived for compliance in the categories:

- < 80 %
- ≥ 80 %

The study treatment exposure (i.e., duration of treatment including interruptions) and study treatment exposure excluding any interruptions will be expressed in weeks for summary tables (i.e., calculated days of exposure are divided by 7), and corresponding categorical variables (not mutually exclusive) are derived (i.e.,  $\geq 24$ ,  $\geq 48$ ,  $\geq 72$ ,  $\geq 96$ ,  $\geq 120$ ,  $\geq 144$  weeks). The number and percent of subjects with 0, 1 or >1 treatment interruptions of >30 days are presented in the exposure table.

Exposure and compliance variables are summarized for the RUBATO OLES, RUBATO pool (SS) (Maci/Maci arm only), and the RUBATO TMAS by means of descriptive statistics (N, mean, standard deviation [SD], median and range [minimum and maximum], and IQ range) for the continuous variables and by means of number and percentage of subjects for categorical variables.

Study drug log data and derived exposure and compliance data will be also listed for the RUBATO OLES and the RUBATO TMAS.

## 5.4. Safety Analysis

The following safety endpoints are defined for analysis:

- Treatment-emergent AEs and SAEs up to 30 days after study treatment discontinuation;
- AEs leading to death;
- AEs leading to premature discontinuation of study treatment;
- AEs of special interest (anemia/hemoglobin decrease, hepatic adverse events of special interest, hypotension, edema and fluid retention) and COVID-19 related AEs. AEs of special interest (AESI) and COVID-19 related AEs are defined using a selection of preferred terms (Internal MedDRA Query). The full definition is included in Section 6.7 Appendix 7;
- (Change in) vital signs (systolic and diastolic arterial BP and pulse rate), including peripheral oxygen saturation (SpO<sub>2</sub>) and body weight over time;
- Treatment-emergent decrease in systolic blood pressure (SBP) up to 30 days after study treatment discontinuation:
- Treatment-emergent marked laboratory abnormalities up to 30 days after study treatment discontinuation;
- (Change in) laboratory parameters over time;
- (Change in) echocardiography parameters over time;
- Treatment-emergent echocardiography abnormalities (valvular defects) up to 30 days after study treatment discontinuation.

For all continuous safety variables, descriptive statistics will include the N, mean, standard deviation [SD], median and range [minimum and maximum] and IQ range. Categorical variables will be summarized using frequency counts and percentages. Unless otherwise specified, data are summarized by the treatment arms defined in Table 3 for the corresponding analysis set.

#### 5.4.1. Adverse Events

An adverse event (AE) is defined as any term reported by the Investigator in the "Adverse Event" eCRF form. The original terms used by the Investigators to describe AEs are assigned preferred terms (PT) and system organ class (SOC) for classification and tabulation using the latest implemented MedDRA version dictionary.

Any AE occurring at or after the study treatment start within the analysis set up to 30 days after the analysis set EOT (limits included) is considered to be treatment-emergent.

The following definitions are relevant for the analysis of the adverse events.

• Frequency of the adverse events

All AEs reported more than once within a subject (as qualified by the same preferred term(s)) are counted once in the frequency table. In the event that the reported AE is assigned to several preferred terms, subjects are counted for each individual preferred term.

### • Intensity of the adverse events

For AEs reported more than once for a subject (as qualified by the same preferred term(s)) but with different intensities, the worst intensity is considered. The categories of intensity are defined as follows: mild, moderate and severe. If intensity is missing, the event is considered severe.

### Relationship of the adverse events

Relationship to study treatment is defined as 'related' (yes) or 'not related' (no). For AEs reported more than once within a subject (as qualified by the same preferred term(s)), the strongest relationship reported (i.e., 'related') is considered. Adverse events with missing relationship are considered in any analysis as related.

• Adverse events leading to discontinuation of study treatment

An AE is defined as leading to discontinuation of study treatment if the corresponding 'Action taken with study treatment' field in the eCRF "AE" form is 'Drug withdrawn'.

• Serious adverse events

A SAE is an AE for which the corresponding 'Serious?' field in the eCRF AE form is ticked 'Yes'. If the information on seriousness is missing, the adverse event is considered serious.

AEs with fatal outcome

An AE is considered having fatal outcome if the tick box "Fatal" for "Outcome" on the eCRF Adverse Event page is checked.

• Adverse events of special interest (AESIs) and COVID-19 related AEs

AEs of special interest are defined using a selection of preferred terms (Internal MedDRA Query) as detailed in Section 6.7 Appendix 7 Adverse Events of Special Interest and COVID-19 related AEs.

• Incidence rate per 100 subject-years of observation (SYO)

In order to account for differences in the time of observation among subjects, for some event types, tables will present the subject-years of observation (SYO) and the incidence rates per 100 subject-years. The subject-observation time will be calculated, for each subject, as follows:

1. For subjects without event of interest: by considering the treatment duration as (EOT date – treatment start date + 1);

2. For subjects with event of interest: by considering the treatment duration up to the start date of first event (min [date of first event, EOT date] – treatment start date + 1)

SYO will be calculated by first summing the subject-observation time for all subjects and then dividing the results by 365.25 days.

The incidence rate for the event of interest, per 100 subject-years, will be calculated by dividing the number of subjects with event of interest by the SYO and multiplying by 100:

Adjusted Incidence Rate =  $100 \times (Number of subjects with at least one event of interest / SYO)$ 

# • Pooling of AEs

For the RUBATO TMAS and RUBATO pool, AEs from DB and OL study are pooled. AEs that started in the DB study and were still ongoing on Day 1 of the OL study are reported in the 'Ongoing Adverse Events from AC-055H301' OL eCRF form. AEs included in the OL eCRF as 'ongoing' from the DB study and the original AEs included in the DB eCRF will be merged using a dedicated ID linking variable included in the related SDTM datasets. If the event worsened in intensity/seriousness after start of study treatment in the OL study, such an event was reported in the usual Adverse Event OL eCRF Form.

The following rules will be used by merging the SDTM datasets:

- The outcome as entered in OL study will be used for the analysis (even if not yet entered due to AE still ongoing)
- o If the action taken for an ongoing AE is given as temporarily interrupted in the DB study database, and the action taken is missing, none, not applicable, or unknown in the OL study database, then the value from the DB will be retained. For all the other cases the action taken as entered in OL study will be used for the analysis

If an event with (partially) missing onset date in the DB study is also entered on the form "Ongoing adverse events from AC-055H301" eCRF page in the OL, this AE will not be considered as treatment-emergent with respect to the OL period (i.e., in subjects of the RUBATO TMAS receiving placebo during DB study), and no dates or other variables will be imputed if missing or partial. Such events will appear in listings only and flagged as DB period event.

All adverse event summary tables described below will be provided for the RUBATO OLES, the RUBATO TMAS, and for the Macitentan 10 mg/Macitentan 10 mg arm of the RUBATO pool (SS), if not otherwise specified.

An overall summary table of AEs will be provided, containing number and percentages of subjects having experienced at least 1 occurrence for the following categories of AEs:

- Treatment-emergent AE
- Treatment-emergent AE related to study treatment

- Treatment-emergent serious AE (SAE)
- Treatment-emergent SAE related to study treatment
- AEs leading to premature discontinuation of study treatment
- Treatment-emergent Fatal (leading to death) AE
- Severe treatment-emergent AE

In order to account for differences in the time of observation among subjects in the RUBATO TMAS, and for the Macitentan 10 mg/Macitentan 10 mg arm of the RUBATO pool (SS), the subject-years of observation (SYO) and the incidence rate per 100 subject-years will be presented for the following categories of AEs:

- Treatment-emergent serious AE (SAE)
- AEs leading to premature discontinuation of study treatment

Separate summary tables (containing number and percentages of subjects) will be provided by SOC and PT within each SOC for the following categories of AEs:

- Treatment-emergent AEs
- Treatment-emergent SAEs
- AEs leading to discontinuation of study treatment
- Treatment-emergent AEs related to study treatment
- Treatment-emergent SAEs related to study treatment
- Treatment-emergent SAEs leading to discontinuation of study treatment
- Treatment-emergent Fatal AEs.

The summary tables are presented in descending order (e.g., SOC and PT within each SOC with the highest number of occurrences appears first). For the summaries on the RUBATO OLES, sorting is done considering the treatment arms in the following sequence: OL Macitentan 10 mg, DB-Macitentan 10 mg, DB-Placebo. In case of equal frequency of different SOC/PTs, alphabetical order is used.

Similarly, separate summary tables (containing number and percentages of subjects) will be provided by PT for the following categories of AEs:

- Treatment-emergent AEs
- Treatment-emergent SAEs
- AEs leading to discontinuation of study treatment
- Treatment-emergent AEs related to study treatment
- Treatment-emergent SAEs related to study treatment

- Treatment-emergent SAEs leading to discontinuation of study treatment
- Treatment-emergent AEs by maximum intensity
- Treatment-emergent AESI, serious AESI, AESI leading to discontinuation of study treatment,
   AESI with fatal outcome
- Treatment-emergent COVID-19 related AEs, serious COVID-19 related AEs, COVID-19 related AEs leading to discontinuation of study treatment, COVID-19 related AEs with a fatal outcome

For each category of AESI, and for COVID-19 related AEs, an overall summary table will be provided, containing number and percentages of subjects having experienced at least 1 occurrence for the following categories: Any AE (plus worst severity of any AE), Any related AE, Any fatal AE, Any SAE, Any related SAE, Any AE leading to discontinuation of study treatment. For the incidence of subjects with any AESI/COVID-19 related AE, this table will also present 95% Clopper-Pearson CL, and the subject-years of observation (SYO) plus incidence rate per 100 subject-years.

In addition to the summary tables, listings will be provided based on the RUBATO pool (SS), displaying:

- AEs
- SAEs
- AEs leading to discontinuation of study treatment
- AEs of special interest
- All AEs in subjects who had any COVID-19 related AE
- All AEs in subjects who had at least one treatment interruption of >30 days. In this listing, AEs with onset date during the interruption(s) are flagged along with the "Day of AE onset relative to last intake prior to treatment interruption" derived as AE start date treatment end date prior to interruption + 1. Only events with a start date during an interruption of >30 days are flagged this way.

For each AE it will be flagged if started in OL or DB period and whether considered treatmentemergent.

#### 5.4.2. Deaths

A summary table will be provided, containing number and percentages of subjects who died on RUBATO pool (SS). Frequencies for the following parameters will be included in the summary table:

- Number of subjects who died
- Primary cause of death

The summary will be based on the "Death" eCRF modules from the DB and the OL eCRF. The summary table is presented by descending order of PT according to the incidence of deaths in the maci/maci treatment arm. The summary will be provided if at least 3 deaths have occurred overall. A corresponding listing is provided and for each death it will be flagged if started in OL or DB period.

## 5.4.3. Vital Signs

Vital signs parameters include systolic and diastolic blood pressure (mmHg), pulse rate (bpm) SpO<sub>2</sub> (%), and body weight (kg) and are summarized by displaying descriptive statistics for the observed values at baseline, for the observed post-baseline assessments, and for the absolute changes from analysis set baseline to each post-baseline visits/timepoint. Except for baseline, only treatment-emergent assessments will be included. Assessments dated after the study treatment start up to 30 days after analysis set EOT (limits included) are considered to be treatment-emergent.

The following nominal visits/timepoints will be displayed for the RUBATO pool (SS):

- DB Baseline ^ ( ~ analysis set baseline)
- DB Week 16
- DB Week 52
- OL Baseline ^
- OL Week 26
- OL Week 52
- OL Week 78
- OL Week 104
- OL Week 130
- OL Week 156

The following nominal visits/timepoints will be displayed for the OLES:

- OL Baseline ^ ( ~ analysis set baseline)
- OL Week 26
- OL Week 52
- OL Week 78
- OL Week 104
- OL Week 130
- OL Week 156

<sup>^</sup> This is not a nominal visit but the derived baseline. In the RUBATO pool (SS), the same assessment may be displayed under 2 timepoints "DB Week 52" and "OL Baseline".

Data is included for analysis regardless of the location (left arm, right arm) or the position of measurement (supine or sitting).

For the RUBATO pool (SS), change from baseline in systolic and diastolic arterial BP, SpO<sub>2</sub> (%) and pulse rate over time will also be graphically presented based on box plots, on a time axis scaled by the target days of nominal visits at DB Week 16, DB Week 52, OL Baseline, OL Week 26, OL Week 52, OL Week 78, OL Week 104. The box indicates the interquartile range, a horizontal line within the box indicates the median, and a diamond shape indicates the mean. Whiskers denote minimum and maximum values within the boundary of +/- 1.5 times the size of the interquartile range. Circles indicate outliers from +/- 1.5 times the size of the interquartile range. A reference line at zero change is drawn.

A decrease in SBP is considered if a post-treatment SBP measurement (scheduled or unscheduled) up to 30 days after analysis set EOT (limits included) is <90 mmHg [or <85 mmHg for adolescents (<18 years old) who are < 150 cm in height] and was not present at baseline. The incidence (number, percentage, and 95% CL using ClopperPearson formula) of subjects with at least one treatment-emergent low systolic blood pressure (SBP) will be summarized for the RUBATO OLES, RUBATO pool (SS) (Maci/Maci arm only), and the RUBATO TMAS. Denominator is the number of subjects with at least one treatment-emergent SBP measurement available. For the RUBATO OLES and the RUBATO pool, the number and percentage of subjects with a decrease in SBP is also summarized by visit.

Blood pressure, pulse rate, SpO<sub>2</sub>, height and body weight measurements will be reported in a subject listing for the RUBATO pool (SS). Position (supine or sitting) and location (left or right arm) for vital signs will be included. Each value will be flagged as assessed during OL or DB period and whether considered treatment-emergent.

### 5.4.4. Laboratory

Safety laboratory samples are centrally analyzed by Covance and the results are electronically transferred into the clinical databases of the two studies. In exceptional cases, the protocols allow the utilization of local laboratories. Local laboratory analysis results are entered in the eCRF. Quantitative results from local laboratories are not summarized (i.e., not included in summary statistics or graphical representations). Qualitative results like (marked) abnormality categorization, liver test elevation categories, etc. are derived from local laboratory data and summarized together with qualitative results derived from central laboratory data. Values from unscheduled visits are not included in by visit/timepoint summaries but are included in the listings and in the summaries for marked abnormalities and liver function test abnormalities.

Data are evaluated in Standard International (SI) units as provided by the central laboratory. In case of local laboratory, values are converted into SI units. The tests converted in SI are available in SDTM for the analysis. All values reported as below or above the limit of detection (e.g., '< 3', '> 100') are substituted with the limit of detection (e.g., '< 3', is substituted by '3') for the purpose of the analysis. The values are listed including the < or > sign.

Safety laboratory data are summarized by displaying descriptive statistics for the observed values at baseline, for the observed post-baseline assessments, and for the absolute changes from analysis set baseline to each post-baseline visit/timepoint. Except for baseline and FU visit, only treatmentemergent assessments will be included. Assessments dated after the study treatment start date up to and including 30 days after analysis set EOT are considered to be treatment-emergent.

The following selected parameters (SI unit) are included in the descriptive statistics summary tables:

- Hematology: Hemoglobin (g/L), Hematocrit (L/L), Leukocyte count (10^9/L), Neutrophils  $(10^9/L)$ , Lymphocytes  $(10^9/L)$ , Platelet count  $(10^9/L)$ .
- Chemistry: Alanine Aminotransferase (U/L), Aspartate Aminotransferase (U/L), Alkaline phosphatase (U/L), Bilirubin (umol/L), Direct bilirubin (umol/L), Gamma glutamyl transpeptidase (U/L), Creatinine (umol/L), Glomerular Filtration Rate, calculated by central laboratory (mL/min/1.73m<sup>2</sup>).

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

Coagulation tests: Prothrombin Time (sec), Prothrombin Intl. Normalized Ratio (ratio).

The following visits/timepoints will be displayed for the RUBATO pool (SS):

- DB Baseline ^ ( ~ analysis set baseline)
- DB Week 16
- DB Week 52
- OL Baseline ^
- OL Week 26
- OL Week 52
- OL Week 78
- OL Week 104
- OL Week 130
- OL Week 156
- Day 30 FU (aminotransferases and hemoglobin only)

The following visits/timepoints will be displayed for the OLES:

- OL Baseline ^ ( ~ analysis set baseline)
- OL Week 26
- OL Week 52
- OL Week 78
- OL Week 104
- OL Week 130

- OL Week 156
- Day 30 FU (aminotransferases and hemoglobin only)

^ This is not a nominal visit but the derived baseline. In the RUBATO pool (SS), the same assessment may be displayed under 2 timepoints "DB Week 52" and "OL Baseline".

Further analyses as described below will be conducted based on the RUBATO pool (SS), and for hematology parameters hemoglobin, hematocrit, leukocytes, platelets and chemistry parameters ALT, AST, Alkaline phosphatase, total bilirubin, creatinine. Only treatment emergent measurements are included:

• The change from baseline over time is presented based on box plots, on a time axis scaled by the target days of nominal visits at DB Week 16, DB Week 52, OL Week 26, OL Week 52, OL Week 78, OL Week 104. The box indicates the interquartile range, a horizontal line within the box indicates the median, and a diamond shape indicates the mean. Whiskers denote minimum and maximum values within the boundary of +/- 1.5 times the size of the interquartile range. Circles indicate outliers from +/- 1.5 times the size of the interquartile range.

All laboratory tests provided by the central and local laboratory will be listed together for the RUBATO pool (SS), including those from unscheduled visits. Marked laboratory abnormalities (MLAs) are flagged accordingly. Each value will be flagged as assessed during OL or DB period and whether considered treatment-emergent.

### **5.4.4.1.** Marked Laboratory Abnormalities

A laboratory test abnormality is defined as any value outside the normal range as provided by the central and local laboratory. The direction of the abnormality (below or above the normal range) is indicated using 'H' and 'L'.

A marked laboratory abnormality (MLA) is defined as any value that fulfills the applicable condition for LL/HH, as provided in Table 6. The marked laboratory abnormalities (MLA) are derived according to the protocol and listed in Table 6 below. More severe marked abnormalities are indicated by LLL/HHH/HHHH, where applicable.

The definitions of marked abnormal values are based mainly on the Common Terminology Criteria for Adverse Events (CTCAE [CTCAE 2010]) grading system and, in specific cases (e.g., lymphocyte levels), are adjusted based on the known pharmacodynamic effect of the study treatment (e.g., LLL threshold for lymphocytes).

All laboratory data are taken into account regardless of whether they correspond to scheduled (per protocol) or unscheduled assessments, and regardless of whether they were analyzed by local or central laboratory.

Treatment-emergent MLAs are all marked laboratory abnormalities occurring after the study treatment start in the analysis set and up to 30 days after analysis set EOT, that were not present at analysis set baseline (see Section 5.1.2.1 for definition) in the same or worse category (considering

the direction of worsening). In other words, the MLAs are evaluated separately for both directions of worsening (e.g., a post-baseline MLA of "HH" is considered treatment-emergent if the baseline is "L" or "LL" or "LLL" (where applicable) or "H", or within normal limits or missing. On the other hand, it is not considered as treatment-emergent if the baseline is "HH" or "HHH" when applicable). In case of missing baseline, an MLA is considered to not have been present at baseline.

**Table 6:** Thresholds for Marked Laboratory Abnormalities

| Parameter (SI unit) | LL | LLL | НН | ннн |
|---|---|---|---|---|
| Hemoglobin (g/L) | < 100 | < 80 | Increase in > 20 | Increase in > 40 g/L above ULN or |
| | | | g/L above ULN or | above baseline (if baseline is above |
| | | | above baseline (if | ULN) |
| | | | baseline is above | |
| | | | ULN) | |
| Hematocrit (L/L) | < 0.28 | < 0.20 | > 0.55 (female) | > 0.65 |
| | (female) | | > 0.60 (male) | |
| | < 0.32 (male) | | | |
| Platelet count (109 /L) | < 75 | < 50 | > 600 | > 999 |
| Eythrocyte count | ND | ND | ND | ND |
| $(10^{12} / L)$ | | | | |
| Leukocyte count (10 <sup>9</sup> | < 3.0 | < 1.9 | > 20.0 | > 100.0 |
| /L) | | | | |
| Lymphocyte (109/L) | ND | < 0.2 | > 4.0 | >20 |
| Neutrophils (10 <sup>9</sup> /L) | < 1.5 | < 1.0 | ND | ND |
| Eosinophils (10 <sup>9</sup> /L) | ND | ND | > 5.0 | ND |
| AST (U/L)* | ND | ND | ≥3 ULN | ≥5 ULN |
| | | | | ≥ 8 ULN (included as HHHH) |
| ALT (U/L)* | ND | ND | ≥3 ULN | ≥5 ULN |
| | | | | ≥ 8 ULN (included as HHHH) |
| Total bilirubin | ND | ND | ≥2 ULN | ≥5 ULN |
| (umol/L) | | | | |
| Alkaline Phosphatase | ND | ND | > 2.5 ULN | > 5 ULN |
| (U/L) | | | | |
| INR* | ND | ND | ≥ 1.5 ULN or | $\geq$ 2.5 ULN or |
| | | | $\geq$ 1.5 × above | $\geq$ 2.5 × above baseline if on |
| | | | baseline if on | anticoagulation |
| | | | anticoagulation | |
| Creatinine (umol/L)* | ND | ND | >1.5 ULN or | > 3 ULN or |
| • | | | $>1.5 \times above$ | >3 × above baseline (if baseline > |
| | | | baseline (if | ULN) |
| | | | baseline > ULN) | · |
| eGFR (mL/min/1.73 | < 60 | < 30 | ND | ND |
| $m^2$ ) | | | | |
| Blood Urea Nitrogen | ND | ND | > 2.5 ULN | > 5 ULN |
| (mmol/L) | | | | |
| Albumin (g/L) | < 30 | < 20 | ND | ND |
| Glucose (mmol/L) | < 3.0 | < 2.2 | > 8.9 | >13.9 |
| Potassium (mmol/L) | < 3.2 | < 3.0 | > 5.5 | > 6.0 |
| Sodium (mmol/L) | ND | < 130 | > 150 | > 155 |
| Calcium (mmol/L) | < 2.0 | < 1.75 | > 2.9 | > 3.1 |
| Triglyceride (mmol/L) | ND | ND | > 3.42 | > 11.4 |
| Cholesterol (mmol/L)* | ND | ND | > 7.75 | > 12.92 |

The above values come from the protocol Table 4 of the protocol.

For each category (i.e., LL, LLL, HH, HHH, HHHH), the number and percentage of subjects with at least one treatment-emergent MLA will be summarized (separately for hematology/coagulation tests and clinical chemistry). Denominator is the number of subjects with at least one treatment-emergent measurement of the corresponding laboratory parameter available. This summary is provided for the RUBATO OLES, RUBATO pool (SS) (Maci/Maci arm only), and the RUBATO TMAS.

# 5.4.4.2. Additional Liver Function Test and Hemoglobin Abnormalities

The following elevated liver test abnormalities are considered:

- ALT or AST  $\geq 3 \times ULN$
- ALT or AST  $\geq$  5 × ULN
- ALT or AST  $\geq 8 \times ULN$
- ALT or AST  $\geq 3 \times$  ULN and total bilirubin  $\geq 2 \times$  ULN (at the same sample date)
- ALT or AST  $\geq$  3 × ULN and total bilirubin  $\geq$  2 × ULN and alkaline phosphatase < 2 × ULN (at the same sample date)
- ALT or AST  $\geq$  3 × ULN and total bilirubin  $\geq$  2 × ULN (at any post-baseline time point up to 30 days after EOT)

The following hemoglobin abnormalities are considered:

- Hemoglobin < 80 g/L
- Hemoglobin  $\geq 80 \text{ g/L}$  and < 100 g/L
- Hemoglobin < 100 g/L.

The highest ALT or AST value and the lowest hemoglobin at any post-baseline time point of assessment up to 30 days after analysis set EOT (limits included) is considered for classification in the categories above.

For each abnormality category, incidence (number, percentage, and 95% CL using Clopper-Pearson formula) of subjects with at least one treatment-emergent abnormality will be summarized. Denominator is the number of subjects with at least one treatment-emergent measurement of any of the corresponding laboratory parameters available. This summary is provided for the RUBATO OLES, RUBATO pool (SS) (Maci/Maci arm only), and the RUBATO TMAS.

<sup>\*</sup> HH and HHH based on CTCAE 2010 v4.03 (CTCAE 2010)

ALT = alanine aminotransferase; AST = aspartate aminotransferase; eGFR = estimated glomerular filtration rate; INR = International Normalized Ratio; NA = not applicable; ND = not defined; SI = international system of units; ULN = upper limit of normal.

For INR, a subject is considered to be on anticoagulation if the subject took antithrombotic agent (ATC codes B01A) and date of INR assessment is on or after start of anticoagulation therapy.

Using the "evaluation of drug-induced serious hepatotoxicity" (eDISH) plots, graphical representations of maximum treatment-emergent ALT (in multiples of ULN) by maximum treatment-emergent total bilirubin (in multiples of ULN) will be produced, to identify potential Hy's Law cases for each subject. The graph will be on a log10 scale for all subjects having assessments > 0.0625 × ULN for both peaks. Two reference lines will be plotted identifying the 2 × ULN for total bilirubin and 3 × ULN for ALT. The normal subjects are on the left lower quadrant, the possible Hy's Law cases appear on the right upper quadrant. The peak is defined as the maximum value from study treatment start up to 30 days after study treatment discontinuation (for the same subjects, not necessarily the peak of ALT occurs at the same time of the peak of total bilirubin). The same plot is provided for parameter AST and both plots are produced for the RUBATO OLES, RUBATO pool (SS) (Maci/Maci arm only), and the RUBATO TMAS.

All chemistry tests provided by the central and local laboratory, including those from unscheduled visits, will be listed separately for subjects with ALT or AST  $\geq$  3 × ULN and total bilirubin  $\geq$  2 × ULN (at any post-baseline time point up to 30 days after EOT) for the RUBATO pool (SS). Each value will be flagged as assessed during OL or DB period and whether considered treatment-emergent.

## 5.4.5. Echocardiography

Numerical echocardiography parameters include single ventricle ejection fraction (%), Fontan circulation stenosis value (%), ventricular outflow to aorta doppler velocity (m/s), vena contracta diameter (mm) and regurgitant orifice (cm²). Single ventricle ejection fraction (%) is summarized by displaying descriptive statistics for the observed values at baseline, for the observed post-baseline assessments, and for the absolute changes from analysis set baseline to each post-baseline visits/timepoint. Except for baseline, only treatment-emergent assessments will be included. Assessments dated after the study treatment start up to 30 days after analysis set EOT (limits included) are considered to be treatment-emergent.

The following nominal visits/timepoints will be displayed for the RUBATO pool (SS):

- DB Baseline ^ ( ~ analysis set baseline)
- DB Week 52
- OL Baseline ^
- OL Week 52
- OL Week 104
- OL Week 156

The following nominal visits/timepoints will be displayed for the OLES:

- OL Baseline ^ ( ~ analysis set baseline)
- OL Week 52
- OL Week 104

#### OL Week 156

^ This is not a nominal visit but the derived baseline. In the RUBATO pool (SS), the same assessment may be displayed under 2 timepoints "DB Week 52" and "OL Baseline".

The following valvular defects are assessed:

- Severe AV valve regurgitation is present where the vena contracta is ≥ 7 mm or the effective regurgitant orifice is ≥ 0.4 cm² in a post-baseline assessment up to 30 days after analysis set EOT, and not present at baseline. In the eCRF, up to two valve regurgitation values may be collected. If both are present in the eCRF, the largest will be considered for the derivation of Severe AV valve regurgitation.
- Presence of **left ventricular outflow obstruction** is confirmed by a pulsed-wave Doppler velocity > 2.5 m/s in a post-baseline assessment up to 30 days after analysis set EOT, and not present at baseline.

For each of the defects, the incidence (number, percentage, and 95% CL using ClopperPearson formula) of subjects with at least one occurrence (scheduled or unscheduled) will be summarized for the RUBATO OLES, RUBATO pool (SS) (Maci/Maci arm only), and the RUBATO TMAS. Denominator is the number of subjects with at least one corresponding treatment-emergent echocardiography measurement available. For the RUBATO OLES and the RUBATO pool, the number and percentage of subjects with valvular defects is also summarized by visit.

Echocardiographic parameters (all numerical and valvular defects) will be reported in a subject listing for the RUBATO pool (SS). Each value will be flagged as assessed during OL or DB period and whether considered treatment-emergent.

### 5.5. Efficacy Analysis

The following efficacy endpoints are assessed:

Cardiopulmonary exercise testing (CPET)

- The change from analysis set baseline to each scheduled time point in peak VO<sub>2</sub>.
- The change from analysis set baseline to each scheduled time point in VO<sub>2</sub> at VAT.

Physical activity measure by Accelerometer (PA-Ac)

• Change from analysis set baseline to each scheduled time point in mean count per minute of daily PA-Ac.

Other endpoints

• Composite endpoint of event related to Fontan-palliated clinical worsening (time to first occurrence of clinical worsening up to analysis set EOS).

• Composite endpoint of events related to Fontan-palliated morbidity (time to first occurrence of morbidity up to analysis set EOS).

No formal hypothesis testing will be performed, as all efficacy analyses are considered exploratory and no inferential analysis is planned for the efficacy variables.

All efficacy endpoints will be analyzed descriptively.

- All assessments (including the unscheduled ones) are considered and re-assigned to the most appropriate visit according to the rules described in Section 5.1.1.
- Listings of all efficacy variable described below will be provided for the RUBATO pool (FAS).
- To investigate the effect of switching from placebo to macitentan 10 mg, some efficacy endpoints are assessed on the RUBATO pool (FAS). Subjects will be analyzed according to the treatment they were randomized to in the RUBATO DB.
- Following 52 weeks of treatment with either placebo or macitentan 10 mg in the DB study, it must be assumed that the two populations will not be similar in terms of baseline characteristics at the start of the OL study. With this limitation acknowledged, specific efficacy endpoints will be analyzed only for the OL study (i.e., on the OLES), overall and split by DB randomized treatment.

# 5.5.1. Cardiopulmonary Exercise Testing (CPET)

Measurements from CPET over time will be displayed at the following analysis visits (see Section 5.1.1 for assignment of assessments to analysis visits, and Section 5.1.2.1 for baseline in analysis set definitions):

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

The following analysis visits/timepoints will be displayed for the RUBATO pool (FAS):

- DB Baseline (~ analysis set baseline)
- DB Week 16
- DB Week 52
- OL Baseline
- OL Week 52
- OL Week 104
- OL Week 156

The following analysis visits/timepoints will be displayed for the OLES:

- OL Baseline (~ analysis set baseline)
- OL Week 52
- OL Week 104

#### • OL Week 156

In the RUBATO pool (FAS), the same assessment may be displayed under 2 timepoints "DB Week 52" and "OL Baseline".

The following endpoints related to CPET are defined:

- Change in peak VO<sub>2</sub> (mL/kg/min), from analysis set baseline to each scheduled time point.
- Change in VO<sub>2</sub> at VAT, from analysis set baseline to each scheduled time point.

Derived as:

Value at scheduled timepoint – Value at analysis set baseline

The values used for peak  $VO_2$  and  $VO_2$  at VAT at baseline and at each scheduled time point above (including the unscheduled ones, within the pre-defined corresponding analysis visits, see Section 5.1.1) will be based on a blinded data evaluation by the independent central reading facility. In case an assessment has been evaluated as "invalid" by the independent central reading facility, it will be ignored.

Baseline peak VO<sub>2</sub> and VO<sub>2</sub> at VAT is not re-derived for the RUBATO pool (FAS) but taken from the RUBATO DB CSR analysis.

For the OLES, baseline peak VO<sub>2</sub> and VO<sub>2</sub> at VAT are derived in a similar manner, i.e., among all available measurements evaluated as "valid" by the central reading facility, the latest assessment prior or at the OL treatment start date (see Section 5.1.2.2) is considered baseline. If no "valid" assessment exists, baseline is imputed with the median value observed at baseline from the remaining subjects (within the DB treatment arm, i.e., DB-placebo or DB-Macitentan 10 mg).

No imputation of missing or invalid post-baseline peak VO<sub>2</sub> and VO<sub>2</sub> at VAT is performed, i.e., data summaries will be based on observed measurements (excluding invalid results).

Peak VO<sub>2</sub> and VO<sub>2</sub> at VAT will be summarized displaying descriptive statistics for the observed values at baseline, for the observed value at each post-baseline assessment, and for the absolute changes from baseline to each post-baseline assessment in analysis sets RUBATO OLES and RUBATO pool (FAS). For the RUBATO pool (FAS), to graphically display changes, a plot of the mean changes (±SE) in peak VO<sub>2</sub> and in in VO<sub>2</sub> at VAT from analysis set baseline over time will be displayed by treatment arm. A reference line is included at zero change and baseline is added to the time axis to visualize an initial change from zero.

In addition, for the RUBATO pool (FAS), Spaghetti plots will be presented by treatment arm to explore the longitudinal pattern of change from baseline in Peak VO<sub>2</sub> and VO<sub>2</sub> at VAT considering all the observed values (from scheduled or unscheduled assessments) and the actual assessment day in RUBATO pool.

Peak VO<sub>2</sub> and VO<sub>2</sub> at VAT will be reported in a subject listing for the RUBATO pool (FAS). Each value will be flagged as assessed during OL or DB period.

### 5.5.2. Physical Activity Measure by Accelerometer

The daily physical activity (counts/min) of the subject is assessed via accelerometer during the daytime. In RUBATO DB, data are collected for 9 consecutive daily daytime periods after Visit 1, after the week 16 visit and before the week 52 visit (which may be selected as baseline for the RUBATO OLES). In RUBATO OL, data are collected for 9 consecutive daily daytime periods after the enrollment visit at Day 1 (mapped to analysis visit "OL Baseline", if available considered baseline for the RUBATO OLES), and after the visits at weeks 26, 52, and 78 visit and before the week 104 visit.

The accelerometry central reading facility will read daily counts/min and will analyze duration of daily activity and time (minutes) which will be transferred to the Sponsor.

For all post baseline assessments during OL period, the 9-day time period is selected by taking the first (in chronological order) interval of 9 consecutive days with at least 4 complete daily time periods within the corresponding time window (i.e., the 9-day time period should not necessarily fall entirely in the corresponding time window, but it should overlap with the time window for at least 1 day). All assessments (including the unscheduled ones) will be mapped based on the Study Day in analysis set (see Section 5.1.1), irrespective of premature study treatment discontinuation before the assessment. To be considered evaluable, physical activity should have been measured for at least 4 complete daily daytime periods (out of 9 consecutive days) at a specific time point of assessment. For the RUBATO pool (FAS), the mean count per minute at analysis visits "DB Baseline", "DB Week 16", and "DB Week 52" is taken from the RUBATO DB ADaM.

To derive baseline mean count per minute of daily PA-Ac for the RUBATO OLES, the PA-Ac data from the OL visit 1 is considered. The 9-day time period is selected by taking the first (in chronological order) interval of 9 consecutive days with at least 4 complete daily time periods, at or after OL treatment start date up to 30 days after OL treatment start. To be considered evaluable, physical activity should have been measured for at least 4 complete daily daytime periods (out of 9 consecutive days) at baseline. A complete day is defined as a record of at least 7 hours of daily daytime data.

The values used for the PA-Ac at baseline and each post-baseline assessment are based on data evaluation by the accelerometry central reading facility.

Mean counts per minute of daily PA-Ac are calculated by dividing the sum of all activity counts (Y axis) collected during wear time for a complete day by the number of minutes of wear time in that day across all valid days (at least 4 days out of 9 days).

The activity counts collected during wear time is identifiable with "WearFilteredAxisYcounts" in Data Transfer Specifications (DTS); the number of minutes of wear time corresponds to the "WearMinutes" variable in DTS.

A complete day is defined as a record of at least 7 hours of daily daytime data, i.e., a complete day if "WearMinutes" >= 7\*60, (after excluding the periods when the device was apparently not worn [Troiano 2008]).

In summary, to compute the mean counts per minute of daily PA-Ac, it is necessary to identify all complete days; if less than 4 complete days out of 9 are identified then value is missing, otherwise, if at least 4 complete days out of 9 are identified, then the value is calculated on the complete days only.

The following endpoint related to PA-Ac are defined:

• change from analysis set baseline to each scheduled time point in mean count per minute of daily PA-Ac from analysis, derived as:

Value at scheduled timepoint – Value at analysis set baseline

Mean count per minute of daily PA-Ac will be summarized displaying descriptive statistics for the observed values at baseline, for the observed value at each post-baseline assessment, and for the absolute changes from baseline to each post-baseline assessment in analysis sets RUBATO OLES and RUBATO pool (FAS). For the RUBATO pool (FAS), to graphically display changes, a plot of the mean changes (±SE) in mean count per minute of daily PA-Ac from analysis set baseline over time will be displayed by treatment arm. A reference line is included at zero change and baseline is added to the time axis to visualize an initial change from zero.

The following analysis visits/timepoints will be displayed for the RUBATO pool (FAS):

- DB Baseline (~ analysis set baseline)
- DB Week 16
- DB Week 52
- OL Baseline
- OL Week 26
- OL Week 52
- OL Week 78
- OL Week 104

The following analysis visits/timepoints will be displayed for the OLES:

- OL Baseline (~ analysis set baseline)
- OL Week 26
- OL Week 52
- OL Week 78
- OL Week 104

In addition, for the RUBATO pool (FAS), spaghetti plots will be presented by treatment arm to explore the longitudinal pattern of change from baseline in mean count per minute of daily PA-Ac considering all the observed values (from scheduled or unscheduled assessments) and the actual assessment day in RUBATO pool.

PA-Ac data will be reported in a subject listing for the RUBATO pool (FAS). Each value will be flagged as assessed during OL or DB period.

## 5.5.3. Fontan-palliated Clinical Worsening and Morbidity Events

The following clinical events endpoints are assessed based on the RUBATO pool (FAS) only:

- Composite endpoint of events related to Fontan-palliated clinical worsening and,
- Composite endpoint of events related to Fontan-palliated morbidity.

The dates of occurrence of each component of the above two clinical events endpoints are reported in the eCRF.

For each composite endpoint, a subject is considered as having an event if the investigator reports the occurrence of any of the individual component in the eCRF (data from RUBATO DB and RUBATO OL are pooled for this purpose), with an event date on or after the date of randomization. Subjects who did not experience an event will be right censored at EOS (as defined in Section 5.1.2.4).

The times to clinical events are expressed in weeks and calculated as:

- For subjects with an event: the earliest date of occurrence of any of the individual components minus date of randomization plus 1 divided by 7,
- For censored subjects: the EOS date minus date of randomization plus 1 divided by 7.

# Composite endpoint of events related to Fontan-palliated clinical worsening

The components of the composite endpoint of events related to Fontan-palliated clinical worsening are the following (these are all assessed by the investigator and recorded in the eCRFs):

- Unscheduled hospitalization for Fontan-palliated morbidity event.
- Signs and symptoms of heart failure, requiring change in diuretic therapy.
- Clinical worsening leading to interventions related to the Fontan-palliated condition.
- Worsening to NYHA FC III, investigator assessed using the Specific Activity Scale.
- Signs and symptoms requiring the addition of a new class of cardiovascular medication (e.g., nitrates, alpha-blockers, or Endothelin receptor antagonists (ERAs)), or insertion of a pacemaker.
- Failing-Fontan defined as one or more of the following:
  - Enlisted on the active list for heart transplantation or effective heart transplantation,

- Reoperation (e.g., mechanical circulatory support, Fontan take down, Fontan revision / conversion, AV valve repair/replacement),
- Worsening to NYHA FC IV, investigator assessed using the Specific Activity Scale,
- Protein-losing enteropathy (PLE),
- Plastic bronchitis/chyloptysis,
- Peritoneal, pleural, mediastinal, or pericardial effusions,
- Severe hepatic impairment,
- Severe renal impairment,
- Death related to Failing-Fontan.

Clinical events are reported in "Clinical worsening events" section of the eCRF.

### Composite endpoint of events related to Fontan-palliated morbidity.

The components of the composite endpoint of events related to Fontan-palliated morbidity are the following:

- Ventricular tachyarrhythmia or supraventricular tachyarrhythmia,
- Thrombotic or hemorrhagic complications (including thromboembolism and hemoptysis).

Clinical events are reported in "Other Fontan-palliated morbidity events" section of the eCRFs.

For each of the two composite endpoints listed above the time to the clinical event will be analyzed, separately, using the Kaplan-Meier (KM) product limit method, providing estimates for each treatment arm and corresponding 95% two-sided CLs at DB weeks 26 and 52, and at OL Weeks 26, 52, 78, 104, 130, 156. The CLs are constructed using Greenwood's formula (Collett 2003) for the standard error of the Kaplan-Meier estimate and are added to the plot. The number of subjects at risk, censored, and with events will be computed and displayed at each time point for each group.

Data will be summarized in tables or figures, including: number of events, number of censored observations, number of subjects at risk, and KM estimates of the survival function for time-to-event variables.

The graph of the estimated survival function of the time to first composite clinical endpoint for each treatment arm obtained from the Kaplan-Meier product-limit method will be displayed up to the time at which at least 10% of all subjects remain at risk of an event. The graphical presentation follows the recommendations from (Pocock 2002).

Individual subject's listings based on the RUBATO pool (FAS) will be provided for both composite endpoints (including details of <u>all</u> (i.e., not only first) individual component events) separately, indicating period (OL or DB period) at time of clinical event.

## 5.6. Other Analyses

## 5.6.1. Definition of Subgroups and subgroup analyses

**Table 7:** Table of Subgroups for Analyses

| Subgroup | Definition |
|---------------------------------|------------------|
| Age (as defined in Section 6.2) | • 12 - <18 years |
| | • ≥ 18 years |

The following analyses are presented by age subgroups in the same way as described above for the overall group:

- Study Disposition (for OLES and TMAS)
- Treatment Disposition (for OLES and TMAS)
- Demographic Characteristics (for OLES and TMAS)
- Baseline Characteristics (for OLES and TMAS)
- Study Treatment Exposure (for RUBATO pool, OLES and TMAS)
- Liver and Hemoglobin Abnormalities (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- Descriptive statistics of vital signs by visit (for RUBATO and OLES)
- Overall summary table of AEs (Any AE, related AE, SAE, related SAE, AE leading to premature discontinuation of study treatment, fatal AE, severe AE) (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- Treatment-emergent AEs by SOC and PT within each SOC (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- Treatment-emergent AEs by PT (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- Treatment-emergent SAEs by SOC and PT within each SOC (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- Treatment-emergent SAEs by PT (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- AEs leading to premature discontinuation of study treatment by SOC and PT within each SOC (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- AEs leading to premature discontinuation of study treatment PT (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- Treatment-emergent AESI by PT (for RUBATO pool Maci/Maci Arm, OLES and TMAS)
- Number of subjects who died and primary cause of death (for RUBATO pool)
#### 6. SUPPORTING DOCUMENTATION

#### 6.1. **Appendix 1: List of Abbreviations**

AΕ Adverse event

AESI Adverse Events of Special Interest

Alanine aminotransferase ALT

ANCOVA Analysis of covariance

> AST Aspartate aminotransferase

ATC Anatomic Therapeutic Chemical

**CPET** Cardiopulmonary Exercise Testing

CLConfidence Limit

Clinical study report CSR

DB Double Blind

DTS **Data Transfer Specifications** 

eCRF Electronic case report form

EOS **End-of-Study** 

EOT **End-of-Treatment** 

FAS Full Analysis Set

FC Functional class

International Council on Harmonisation **ICH** 

LV Left ventricle

MAR Missing at random

MedDRA Medical Dictionary for Regulatory Activities

NT-pro-BNP n-terminal pro-brain natriuretic peptide

NYHA New York Heart Association

OL Open Label

**OLES** Open-label Extension analysis set

PA-Ac Physical Activity measured by Accelerometer

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

PD Protocol deviation

PT Preferred Term

QTL Quality Tolerance Limit

Right ventricle RV

Serious adverse event SAE

SAP Statistical analysis plan

SE Standard Error

| SD | Standard Deviation |
|---|---|
| SDTM | Study Data Tabulation Model |
| SI | International system of units |
| SMQ | Standardised MedDRA Query |
| SOC | System organ class |
| $SpO_2$ | Peripheral oxygen saturation |
| SS | Safety Analysis Set |
| TCPC | Total cavopulmonary connection |
| TMAS | Total Macitentan analysis set |
| ULN | Upper limit of normal |
| VAT | Ventilatory anaerobic threshold |
| $VO_2$ | Oxygen uptake/consumption $[\dot{V}O_2 \text{ is a flow} = \text{a ratio of Volume of Oxygen by unit of time}]$ |
| WHO | World Health Organization |

# 6.2. Appendix 2: Changes to Protocol-Planned Analyses

This study was prematurely discontinued by the sponsor. Study results will be presented in an abbreviated CSR.

While all safety data obtained will be summarized, only a subset of the protocol-specified efficacy endpoints and none of the protocol-specified pharmacoeconomic endpoints will be summarized. Due to the early termination of this long-term study, only key safety data (SAE, AEs leading to discontinuation, AESI) are presented adjusted for subject-years of observation. Subgroup analyses are limited to analyses by age-group.

# 6.3. Appendix 3: Demographic and Baseline Characteristics

# 6.3.1. Demographics

Demographic data will be presented for the RUBATO OLES and the RUBATO TMAS.

Weight, Height, Body Mass Index (BMI) will be taken/derived from the analysis set baseline.

Age and sex are collected on the RUBATO OL study Demographics page and used for the RUBATO OLES and for RUBATO TMAS subjects from the placebo arm in the RUBATO DB SS. For RUBATO TMAS subjects from the macitentan arm in the RUBATO DB SS, the RUBATO DB demographics page is used.

All other demographic variables are taken from the RUBATO DB demographics page.

Table 8 presents a list of the demographic variables that will be summarized RUBATO OLES and the RUBATO TMAS. Demographics will also be summarized by subgroups as defined in Section 5.6.1.

**Table 8:** Demographic Variables

| Continuous Variables: | Summary Type |
|---|---|
| Age | Descriptive statistics (N, mean, |
| Weight (kg) | standard deviation [SD], median |
| Height (cm) | and range [minimum and |
| Body Mass Index (BMI) (kg/m²) | maximum], and IQ range). |
| Categorical Variables | |
| Age (12–<18, 18–<30, 30–<40, 40-<65, >= 65) | |
| Sex (male, female) | |
| Race (American Indian or Alaska Native, Asian, Black or African | |
| American, Native Hawaiian or other Pacific Islander, White, Other, Not | |
| Applicable) | Frequency distribution with the |
| Ethnicity (Hispanic or Latino, not Hispanic or Latino, Unknown) | number and percentage of subjects |
| Geographical region (America, Europe, Asia, Oceania) | in each category. |
| Region (US, Non-US) | |
| BMI ([underweight <18.5 kg/m², normal 18.5-<25 kg/m², overweight 25- | |
| <30 kg/m², obese class I 30-<35 kg/m², obese class II 35-<40 kg/m², obese | |
| class III $\geq 40 \text{ kg/m}^2$ ]) <sup>a</sup> | |

<sup>&</sup>lt;sup>a</sup> Body Mass index BMI (kg/m²) is calculated in the eCRF for RUBATO DB, for RUBATO OL, it is derived as Weight (kg) / [Height (cm) / 100]², rounded to one decimal as done in DB eCRF. For adolescents (boys or girls) between 12 and 18 years, BMI-for-age reference equivalent to BMI cutoffs for adults are calculated as provided in Attachment 1 of the RUBATO DB CSR SAP (EDMS-RIM-264216, 1.0).

All demographic data will be reported in subject listings on the RUBATO OLES and the RUBATO TMAS.

#### 6.3.2. Baseline Disease Characteristics

Table 9 presents a list of baseline disease characteristics variables that will be summarized RUBATO OLES and the RUBATO TMAS.

**Table 9:** Baseline Disease Characteristics

| Continuous Variables: | Summary Type |
|---|---|
| Time since Fontan palliation completion (years) at treatment start in analysis set | |
| Peak VO <sub>2</sub> (mL/kg/min) at baseline at analysis set baseline | Descriptive statistics (N, mean, |
| VO <sub>2</sub> at VAT at baseline at analysis set baseline | standard deviation [SD], median and range [minimum and |
| Mean count per minute of daily Physical Activity at baseline at analysis set baseline | maximum], and IQ range). |
| NT-proBNP (pmol/L) at analysis set baseline | |
| Categorical Variables | |
| Congenital heart defect leading to Fontan-palliation as recorded at DB study entry | |
| Dominant ventricular morphology (left and right/mixed) as recorded at DB study entry | |
| Staged reconstructive surgeries performed before completion of the Fontan circulation as recorded at DB study entry | |
| Type of primary TCPC Fontan completion as recorded at DB study entry | Frequency distribution with the |
| Type of secondary TCPC Fontan completion (TCPC=total cavopulmonary connection) as recorded at DB study entry | number and percentage of subjects in each category. |
| Fenestration Status as recorded at DB study entry | |
| PAH specific therapies concomitant at start of study treatment in analysis set | |
| NYHA FC at analysis set baseline | |

# PAH specific therapies concomitant at start of study treatment in analysis set

• PAH specific medications concomitant at start of study treatment in analysis set (see Section 6.5.3 for definition). Pulmonary hypertension specific medications are: sildenafil, sildenafil citrate, tadalafil, vardenafil, udenafil, iloprost, beraprost, epoprostenol, treprostinil, selexipag, bosentan, ambrisentan, riociguat.

All other variables that are presented, are based on data recorded at entry into study RUBATO DB will be derived as described in the RUBATO DB CSR SAP. The remaining variables are re-derived in the same manner as described in the RUBATO DB CSR SAP, based on the analysis set baseline (as defined in Section 5.1.2.1).

All baseline disease characteristics variables will be reported in subject listings on the RUBATO OLES and the RUBATO TMAS.

# 6.4. Appendix 4: Protocol Deviations and Quality Tolerance Limits (QTL)

The description of each protocol deviation (PD) is agreed in the sponsor protocol deviation code list (PD list Version 3, dated 20-Apr-2021). According to this document, each PD is classified as important or not important. A further categorization into one of the following categories is documented in Table 10: Entered but did not satisfy criteria, Developed withdrawal/interruption criteria but not withdrawn/interrupted, Received a disallowed concomitant treatment, Received wrong treatment or incorrect dose, Other.

Only important (i.e., major) protocol deviations will be summarized by category, displaying counts and percentages of subjects with at least one PD within each category for the RUBATO OLES. A separate similar summary of important PDs will be provided by geographical region and site. These summaries are provided for all important (i.e., major) PDs and separately for all COVID-19 related important (i.e., major) PDs.

All reported PDs and all reported COVID-19 related PDs will be reported in subject listings. Both listings are provided for the RUBATO OLES, with important PDs flagged accordingly.

Table 10: PD Classification Based on AC-055H302 (RUBATO OL)

| Condition | Identifier | Important | Categorization of PD for reporting |
|---|---|---|---|
| Subject not enrolled but received study drug | PD_MM.101 | Yes | Received wrong treatment or incorrect dose |
| Informed consent not personally signed and dated by subject /legal representative | PD_MM.102 | Yes | Other |
| Study assessments were performed but no informed consent was signed and dated by subject/legal representative. | PD_MM.103 | Yes | Other |
| Informed consent process (including re-consenting) not followed | PD_MM.104 | Yes | Other |
| Subject enrolled but did not complete Week 52 of RUBATO DB | PD_MM.132 | Yes | Entered but did not satisfy criteria |
| Woman of childbearing potential who did not have a negative serum pregnancy test prior to first intake of OL study drug | PD_MM.133 | Yes | Entered but did not satisfy criteria |
| Other violation before enrollment not listed above | PD_MM.105 | No | Other |
| Woman of childbearing potential who did not agree to perform monthly pregnancy tests up to the end of the S-FU period | PD_MM.134 | Yes | Entered but did not satisfy criteria |
| Woman of childbearing potential who did not agree to use reliable contraception from enrollment and up to at least 30 days after study drug discontinuation | PD_MM.135 | Yes | Entered but did not satisfy criteria |
| Clinical worsening leading to medical interventions including reoperation of Fontan circulation during the enrollment period | PD_MM.136 | Yes | Entered but did not satisfy criteria |
| Systolic BP < 90 mmHg (< 85 mmHg for subjects < 18 years old and < 150 cm of height) at rest | PD_PM.325 | Yes | Entered but did not satisfy criteria |
| Hemoglobin < 75% of the lower limit of normal assessed by central laboratory at enrollment | PD_PM.326 | Yes | Entered but did not satisfy criteria |
| Known or suspected pulmonary veno-occlusive disease | PD_MM.137 | Yes | Entered but did not satisfy criteria |
| Known and documented severe hepatic impairment defined as Child-Pugh Score C | PD_MM.138 | Yes | Entered but did not satisfy criteria |
| Serum AST and/or ALT > 3 x upper limit of normal range assessed by central laboratory at enrollment | PD_PM.327 | Yes | Entered but did not satisfy criteria |
| Severe renal impairment (estimated creatinine clearance < 30 mL/min/1.73m2) assessed by central laboratory at enrollment | PD_PM.328 | Yes | Entered but did not satisfy criteria |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Condition | Identifier | Important | Categorization of PD for reporting |
|---|---|---|---|
| Hypersensitivity to any active substance or excipient of any of the study drugs | PD_MM.139 | Yes | Entered but did not satisfy criteria |
| Treatment with a strong cytochrome P450 3A4 (CYP3A4) inducer within 1 month prior to enrollment (Visit 1) | PD_MM.140 | Yes | Entered but did not satisfy criteria |
| Treatment with a strong CYP3A4 inhibitor within 1 month prior to enrollment (Visit 1) | PD_MM.141 | Yes | Entered but did not satisfy criteria |
| Treatment with a moderate dual CYP3A4/CYP2C9 inhibitor (e.g., fluconazole, amiodarone) or co-administration of a combination of moderate CYP3A4 and moderate CYP2C9 inhibitors within 1 | PD_MM.142 | Yes | Entered but did not satisfy criteria |
| month prior to enrollment (Visit 1) Any factor or condition likely to affect protocol compliance of the | PD MM.143 | Yes | Entered but did not satisfy |
| subject, as judged by the investigator Treatment with another investigational therapy during the OL | PD_MM.144 | Yes | criteria Entered but did not satisfy |
| study Treatment with ERAs other than macitentan | PD_MM.145 | Yes | criteria Entered but did not satisfy criteria |
| Known drug or substance (e.g., alcohol) abuse, unstable psychiatric illness, or any other condition that, in the opinion of | PD_MM.146 | Yes | Entered but did not satisfy criteria |
| the investigator, may interfere with participation in the study Any planned surgical intervention (e.g., organ transplant) during the study period, except minor interventions (e.g., tooth extraction) | PD_MM.147 | Yes | Entered but did not satisfy criteria |
| Any known factor or disease that may interfere with treatment compliance or full participation in the study (e.g., chemotherapy treatment for cancer) or illness with an anticipated life expectancy of less than 12 months. | PD_MM.148 | Yes | Entered but did not satisfy criteria |
| PA-Ac device not correctly assigned or initiated at enrollment | PD_MM.149 | Yes | Other |
| Subject not contacted to remind them to wear PA-Ac device | PD_MM.150 | No | Other |
| Enrollment assessment not done/missing | PD_PP.202 | Yes | Other |
| Pregnancy testing at enrollment not done | PD_PM.301 | Yes | Other |
| Entry enrollment labs are > 4 weeks after EOT Visit in AC-055H301 RUBATO DB | PD_PM.302 | Yes | Other |
| Study drug not withheld prior to assessments at enrollment visit | PD_MM.106 | No | Other |
| CPET at Visit 1 conducted under different conditions than during the AC-055H301 RUBATO DB study | PD_MM.107 | No | Other |
| CPET at Visit 1 done, but not valid/questionable on review by central reading facility | PD_MM.108 | No | Other |
| CPET at Visit 1 not done according to guidelines and central reader manual | PD_MM.109 | No | Other |
| CPET at Visit 1 not done (but required) | PD_MM.151 | No | Other |
| SAE not reported within 24 hours of knowledge, or not reported as per protocol | PD_MM.110 | Yes | Other |
| Other violation at enrollment not listed above | PD_MM.111 | No | Other |
| Subject has no post-baseline safety assessment | PD_PM.303 | Yes | Other |
| Subject has no post-baseline efficacy assessment | PD_PM.304 | Yes | Other |
| PA-AC device not returned/device lost/issues with upload | PD_MM.152 | No | Other |

| Condition | Identifier | Important | Categorization of PD for reporting |
|---|---|---|---|
| Subject does not have sufficient PA-Ac baseline data | PD_PM.305 | No | Other |
| Visit 2 assessment not done/missing | PD_PP.203 | Yes | Other |
| Visit 2 vital signs assessed under different conditions than at baseline | PD_MM.116 | No | Other |
| Visit 2 labs missing/incomplete | PD_PM.306 | Yes | Other |
| Study drug not withheld prior to assessments at Visit 2 | PD_MM.117 | No | Other |
| PA-Ac device not correctly assigned or initiated at Visit 2 | PD_MM.153 | No | Other |
| Subject does not have sufficient PA-Ac data at Visit 2 | PD_PM.329 | No | Other |
| Subject not contacted to remind them to wear PA-Ac device | PD_MM.154 | No | Other |
| PA-Ac device not returned/lost device/upload problems | PD_MM.155 | No | Other |
| CPET at Visit 3 conducted under different conditions than at baseline | PD_PM.307 | No | Other |
| CPET at Visit 3 done, but not valid/questionable on review by central reading facility | PD_PM.308 | No | Other |
| CPET at Visit 3 not done according to guidelines and central reader manual | PD_MM.118 | No | Other |
| CPET at Visit 3 not done | PD_PP.204 | No | Other |
| Visit 3 assessment not done/missing | PD_PP.205 | Yes | Other |
| Visit 3 vital signs assessed under different conditions than at baseline | PD_MM.119 | No | Other |
| Subject does not have sufficient PA-Ac data at Visit 3 | PD_PM.309 | No | Other |
| Visit 3 labs missing/incomplete | PD_PM.310 | Yes | Other |
| Study drug not withheld prior to assessments at Visit 3 | PD_MM.120 | No | Other |
| Visit 4 assessment not done/missing | PD_PP.206 | Yes | Other |
| Visit 4 vital signs assessed under different conditions than at baseline | PD_MM.121 | No | Other |
| Subject does not have sufficient PA-Ac data at Visit 4 | PD_PM.311 | No | Other |
| Visit 4 labs missing/incomplete | PD_PM.312 | Yes | Other |
| Study drug not withheld prior to assessments at Visit 4 | PD_MM.122 | No | Other |
| Visit 5 assessment not done/missing | PD_PP.207 | Yes | Other |
| CPET at Visit 5 conducted under different conditions than at baseline | PD_PM.313 | No | Other |
| CPET at Visit 5 done, but not valid/questionable on review by central reading facility | PD_MM.123 | No | Other |
| CPET at Visit 5 not done according to guidelines and central reader | PD_MM.124 | No | Other |
| manual CPET at Visit 5 not done | PD_PP.208 | No | Other |
| Visit 5 vital signs assessed under different conditions than at baseline | PD_MM.125 | No | Other |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Condition | Identifier | Important | Categorization of PD for reporting |
|---|---|---|---|
| Subject does not have sufficient PA-Ac data at Visit 5 | PD_PM.314 | No | Other |
| Visit 5 labs missing/incomplete | PD_PM.315 | Yes | Other |
| Study drug not withheld prior to assessments at Visit 5 | PD_MM.126 | No | Other |
| Visit 6 assessment not done/missing | PD_PP.214 | Yes | Other |
| Visit 6 vital signs assessed under different conditions than at baseline | PD_MM.171 | No | Other |
| Visit 6 labs missing/incomplete | PD_PM.332 | Yes | Other |
| Study drug not withheld prior to assessments at Visit 6 | PD_MM.172 | No | Other |
| Visit 7 assessment not done/missing | PD_PP.215 | Yes | Other |
| CPET at Visit 7 conducted under different conditions than at baseline | PD_PM.333 | No | Other |
| CPET at Visit 7 done, but not valid/questionable on review by central reading facility | PD_MM.173 | No | Other |
| CPET at Visit 7 not done according to guidelines and central reader manual | PD_MM.174 | No | Other |
| CPET at Visit 7 not done | PD_PP.216 | No | Other |
| Visit 7 vital signs assessed under different conditions than at baseline | PD_MM.175 | No | Other |
| Visit 7 labs missing/incomplete | PD_PM.334 | Yes | Other |
| Study drug not withheld prior to assessments at Visit 7 | PD_MM.176 | No | Other |
| Visit 8 assessment not done/missing | PD_PP.217 | Yes | Other |
| Visit 8 vital signs assessed under different conditions than at baseline | PD_MM.177 | No | Other |
| Visit 8 labs missing/incomplete | PD_PM.335 | Yes | Other |
| Study drug not withheld prior to assessments at Visit 8 | PD_MM.178 | No | Other |
| Visit 9 assessment not done/missing | PD_PP.218 | Yes | Other |
| CPET at Visit 9 conducted under different conditions than at baseline | PD_PM.336 | No | Other |
| CPET at Visit 9 done, but not valid/questionable on review by central reading facility | PD_MM.179 | No | Other |
| CPET at Visit 9 not done according to guidelines and central reader manual | PD_MM.180 | No | Other |
| CPET at Visit 9 not done | PD_PP.219 | No | Other |
| Visit 9 vital signs assessed under different conditions than at baseline | PD_MM.181 | No | Other |
| Visit 9 labs missing/incomplete | PD_PM.337 | Yes | Other |
| Study drug not withheld prior to assessments at Visit 9 | PD_MM.182 | No | Other |
| Initiation of forbidden medication | PD_PM.338 | Yes | Received a disallowed concomitant treatment |
| Aminotransferase elevation ≥ 3 x ULN and study drug not interrupted or discontinued | PD_PM.316 | Yes | Developed<br>withdrawal/interruption |

| Condition | Identifier | Important | Categorization of PD for reporting |
|---|---|---|---|
| | | | criteria but not |
| | | | withdrawn/interrupted |
| Aminotransferase elevation ≥ 3 x ULN and retests not done per protocol | PD_PM.317 | Yes | Other |
| Hemoglobin < 100 g/L with a decrease from baseline of ≥ 50 g/L and retest not done per protocol | PD_PM.318 | Yes | Other |
| Hemoglobin < 80 g/L with no underlying blood loss and study | PD_PM.319 | Yes | Developed |
| treatment not interrupted | | | withdrawal/interruption<br>criteria but not<br>withdrawn/interrupted |
| Re-introduction of treatment before a) Aminotransferases | PD_PM.320 | Yes | Developed |
| returned to pre-treatment or normal range b) Hemoglobin returned to pre-treatment or normal range | 1 B_1 1111320 | 103 | withdrawal/interruption<br>criteria but not<br>withdrawn/interrupted |
| Blood pressure dropped < 90 mm Hg (< 85 mm Hg for subjects < | PD_PM.321 | Yes | Developed |
| 18 years old and < 150 cm of height and study drug not interrupted | | | withdrawal/interruption<br>criteria but not |
| Subject got progrant during the treatment period or within 20 | PD PM.322 | Voc | withdrawn/interrupted Other |
| Subject got pregnant during the treatment period or within 30 days after treatment discontinuation | PD_PIVI.322 | Yes | Other |
| Subject got pregnant and study drug was not interrupted | PD_PM.330 | Yes | Developed withdrawal/interruption |
| | | | criteria but not |
| Woman of childbearing potential not using reliable contraception | PD_PM.323 | Yes | withdrawn/interrupted<br>Other |
| Pregnancy test was missed | PD_MM.156 | Yes | Other |
| CPET performed out of window of last QA (> 213 days since last QA) | PD_MM.127 | No | Other |
| ECHOC not performed according to guidelines | PD_MM.128 | No | Other |
| Subject received treatment which was not approved for use | PD_MM.157 | Yes | Other |
| Study treatment compliance between 2 visits < 80% or > 120% | PD_PM.324 | Yes | Received wrong treatment or incorrect dose |
| Overall study treatment compliance for the whole treatment | PD_MM.158 | Yes | Received wrong treatment |
| period < 80% or > 120% | _ | | or incorrect dose |
| Study treatment compliance based on subject's report | PD_MM.183 | No | Received wrong treatment or incorrect dose |
| Study medication not stored correctly but subject continued to use it | PD_MM.129 | Yes | Received wrong treatment<br>or incorrect dose |
| Study treatment not administered as per protocol (any dose of | PD MM.159 | Yes | Received wrong treatment |
| study treatment higher than the planned total daily dose in a single day will be considered an overdose) | _ | | or incorrect dose |
| Subject treatment not discontinued although subject (legally | PD_MM.160 | Yes | Developed |
| acceptable representative) decided not to continue treatment | | | withdrawal/interruption criteria but not |
| Cubicat modication and discontinued although in cations | DD 1414464 | V | withdrawn/interrupted |
| Subject medication not discontinued although investigator considers that the subject should not continue treatment | PD_MM.161 | Yes | Developed withdrawal/interruption criteria but not |
| | | | withdrawn/interrupted |
| Sponsor decision to withdraw subject or terminate study and subject was not discontinued within the time indicated by the | PD_MM.162 | Yes | Developed<br>withdrawal/interruption |
| sponsor | | | criteria but not withdrawn/interrupted |

| Condition | Identifier | Important | Categorization of PD for reporting |
|---|---|---|---|
| Visit 2 performed out of window (Day 183 ± 7 days) | PD_PP.209 | No | Other |
| Visit 3 performed out of window (Day 365 ± 7 days) | PD_PP.210 | No | Other |
| Visit 4 performed out of window (Day 547 ± 7 days) | PD_PP.211 | No | Other |
| Visit 5 performed out of window (Day 729 ± 7 days) | PD_PP.212 | No | Other |
| Visit 6 performed out of window (Day 911 ± 7 days) | PD_PP.220 | No | Other |
| Visit 7 performed out of window (Day 1093 ± 7 days) | PD_PP.221 | No | Other |
| Visit 8 performed out of window (Day 1275 ± 7 days) | PD_PP.222 | No | Other |
| Visit 9 performed out of window (Day 1457 ± 7 days) | PD_PP.223 | No | Other |
| Visit EOS performed out of window (EOS + 30-35 days) | PD_PP.213 | No | Other |
| 6-monthly visit performed out of window | PD_MM.163 | No | Other |
| FU-visit performed out of window | PD_MM.164 | No | Other |
| Visit was performed remotely/partly remotely | PD_MM.165 | No | Other |
| SAE not reported within 24 hours of knowledge, or not reported as per protocol | PD_MM.130 | Yes | Other |
| CPET data not sent to central reading facility within 5 working days | PD_MM.166 | No | Other |
| Monthly lab performed out of window | PD_PM.331 | No | Other |
| Monthly lab sample missing | PD_MM.167 | Yes | Other |
| Consecutive lab samples missing/not available without replacement/local labs being done | PD_MM.168 | Yes | Other |
| Oversampling during lab assessments | PD_MM.169 | Yes | Other |
| Lab report not signed within 5 days of receipt | PD_MM.170 | No | Other |
| Other violation during treatment period and follow-up not listed above | PD_MM.131 | No | Other |

During the course of this long-term safety study, two quality tolerance criteria were defined as shown in table 11 below. Both are related to participants' safety.

Table 11: Quality Tolerance Limits as per Integrated Analytical Risk-Based Monitoring Plan

| Critical to Quality Factor | Parameter | Primary Threshold | Captured in PD/PD category |
|---|---|---|---|
| Subjects who meet at least one of<br>the study specific discontinuation<br>criteria must be permanently<br>discontinued. | % subjects not discontinued according to protocol safety criteria. | 10% subjects not discontinued according to protocol safety criteria. Special attention in the first 6 months of treatment (because of placebo roll over patients) | Developed withdrawal/interruption criteria but not withdrawn/interrupted |
| Safety laboratory must be done per time and events schedule in the protocol. | % of subjects with 2<br>missing consecutive safety<br>lab tests and % of missing<br>safety lab test. | 10 % of subjects with 2 missing consecutive safety lab tests | PD_MM.168 |

### 6.5. Appendix 5: Prior and Concomitant Medications

All therapies as collected in the "Previous/Concomitant Medication" eCRF form of the two studies RUBATO DB and RUBATO OL will be pooled for the RUBATO OLES and the RUBATO TMAS.

The original terms used by the investigators to describe therapies are assigned preferred terms for classification and tabulation using the latest version of the World Health Organization (WHO) Drug code and Anatomic Therapeutic Chemical (ATC) class code dictionaries.

# 6.5.1. Prior Medications

Prior medications are defined as any therapy with an end date prior to the date of first intake of study medication in the analysis set.

If the end date is missing and the start date is prior to the date of first intake of study medication in the analysis set, and

- the checkbox for the question 'Ongoing at start of treatment?' is ticked 'No' on the RUBATO DB eCRF form, then the therapy is considered as previous for all subjects in the RUBATO OLES and the RUBATO TMAS.
- the checkbox for the question 'Ongoing at start of treatment?' is ticked 'No' on the RUBATO OL eCRF form, then the therapy is considered as previous in the RUBATO OLES for all subjects and in the RUBATO TMAS for subjects from the placebo arm in the RUBATO DB (SS). In the RUBATO TMAS it is considered concomitant for subjects from the macitentan arm in the RUBATO DB (SS) unless the same record (i.e., same therapy, same start date, missing end date, 'Ongoing at start of treatment?' ticked 'No') is also documented in the DB eCRF. In this case it is also considered previous for the RUBATO TMAS.

#### 6.5.2. Concomitant Medications

Concomitant medications are all therapies that are ongoing at, and/or initiated before date of first intake of study medication in the analysis set and terminated after the date of first intake of study medication in the analysis set, or initiated on or after the date of first intake of study medication in the analysis set up to the date of EOT in the analysis set.

Number and percentages of subjects having taken at least one medication will be presented by Anatomic Therapeutic Chemical (ATC) class (level 4) and PT within each ATC class for the RUBATO OLES and the RUBATO TMAS. All summaries will be tabulated by ATC class, and individual preferred terms within each ATC class. ATC classes will be sorted by descending order. For the summaries on the RUBATO OLES, sorting is done considering the arms in the following sequence: OL Macitentan 10 mg, DB-Macitentan 10 mg, DB-Placebo. If the frequencies of ATC class are the same, alphabetical order will be used. The same rule applies for preferred terms within ATC class.

Subjects who took the same medication more than once (as qualified by the same PT(s)) are counted only once. In case the reported medication is assigned to several PTs, subjects are counted for each individual PT.

All medications will be reported in a subject listing including all subjects with flags to identify prior and concomitant medications accordingly, on the RUBATO OLES and the RUBATO TMAS. This listing is repeated in the subset of subjects who had any COVID-19 related AE.

# 6.5.3. Concomitant Medications at Start of Study Treatment in Analysis Set

Concomitant therapies at start of treatment in analysis set is any treatment that is either ongoing at the start of study treatment or is initiated at the start date of study treatment, identified as follows:

- 'Ongoing at start of treatment? = Yes' ticked by the investigator in the eCRF\*,
   or
- Start date before or on analysis set treatment start date and end date on or after treatment start date,

or

- Start date before or on analysis set treatment start date and end date missing with 'Ongoing at start of treatment?'  $\neq No$ ' in the eCRF\*.
  - \* Based on the RUBATO OL "Previous/Concomitant Medication" eCRF form for OLES and for RUBATO TMAS subjects from the placebo arm in the RUBATO DB SS. Based on the RUBATO DB "Previous/Concomitant Medication" eCRF form for RUBATO TMAS subjects from the macitentan arm in the RUBATO DB SS.

# 6.6. Appendix 6: Intervention Compliance

Not applicable. Only percentage of days with study treatment exposure (excluding interruptions) of the duration of exposure (including interruptions) are reported as described in Section 5.3.

# 6.7. Appendix 7: Adverse Events of Special Interest and COVID-19 related AEs

Adverse events of special interest are defined as follows:

# I. Hepatic events of special interest

AEs are included in this grouping if their coded PTs are included in the "Hepatic disorders" SMQ with including all its sub-SMQ with the exception of "Liver-related coagulation and bleeding disturbances (SMQ)".

### II. Edema and fluid retention

AEs are included in this subgroup if their coded PTs is "Pulmonary congestion" or if within the SMQ "Haemodynamic oedema, effusions and fluid overload (SMQ)" with the exception of PTs containing "site".

# III. Anemia / hemoglobin decrease

AEs are included in this grouping if their coded PTs are included in the SMQs "Haematopoietic erythropenia" OR "Haematopoietic cytopenias affecting more than one type of blood cell (SMQ)" (with the exception of two unspecific PTs: "blood disorder", "blood count abnormal") OR an event with any MedDRA PT containing the text "anaemia".

# IV. Hypotension

AEs are included in this grouping if their coded PTs are: Blood pressure ambulatory decreased, Blood pressure decreased, Blood pressure diastolic decreased, Blood pressure immeasurable, Blood pressure orthostatic decreased, Blood pressure systolic decreased, Blood pressure systolic inspiratory decreased, CT hypotension complex, Diastolic hypotension, Hypotension, Mean arterial pressure decreased, Neonatal hypotension, Orthostatic hypotension, Procedural hypotension, Dialysis hypotension, Hypotensive crisis, Post procedural hypotension.

### **List of COVID-19 related AEs**

AEs are considered as COVID-19 related if their coded PTs are: Asymptomatic COVID-19, Congenital COVID-19, Coronavirus infection, Coronavirus test positive, COVID-19, COVID-19 immunisation, COVID-19 pneumonia, COVID-19 prophylaxis, COVID-19 treatment, Exposure to SARS-CoV-2, Multisystem inflammatory syndrome in children, Occupational exposure to SARS-CoV-2, Post-acute COVID-19 syndrome, SARS-CoV-2 antibody test positive, SARS-CoV-2 carrier, SARS-CoV-2 RNA decreased, SARS-CoV-2 RNA fluctuation, SARS-CoV-2 RNA increased, SARS-CoV-2 sepsis, SARS-CoV-2 test false negative, SARS-CoV-2 test positive, SARS-CoV-2 viraemia, Suspected COVID-19, Vaccine derived SARS-CoV-2 infection, Antiviral prophylaxis, Antiviral treatment, Coronavirus test, Coronavirus test negative, COVID-19 screening, Exposure to communicable disease, Pneumonia viral, SARS-CoV-2 antibody test, SARS-CoV-2 antibody test negative, SARS-CoV-2 RNA undetectable, SARS-CoV-2 test, SARS-CoV-2 test false positive, SARS-CoV-2 test negative.

# 7. REFERENCES

- (CTCAE 2010) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 Published: May 28, 2009 (v4.03: June 14, 2010) U.S. Department of Health And Human Services. National Institutes of Health National Cancer Institute.
- (Collett 2003) Modelling Survival Data in Medical Research, 2nd Edition. Chapman & Hall; 2003.
- (Pocock 2002) Pocock SJ, Clayton TC, G Altman DG. Survival plots of time-to-event outcomes in clinical trials: good practice and pitfalls. Lancet. 2002;359:1686–89.
- (Troiano 2008) Troiano RP, Berrigan D, Dodd KW, Mâsse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008;40(1):181-8.